CLINICAL TRIAL: NCT02942004
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of SAGE-547 Injection in the Treatment of Adult Female Subjects With Severe Postpartum Depression and Adult Female Subjects With Moderate Postpartum Depression
Brief Title: A Study to Evaluate Efficacy and Safety of SAGE-547 in Participants With Severe Postpartum Depression (547-PPD-202B)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 547-PPD-202 B
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Depression
Keywords: Severe Postpartum Depression; SAGE-547
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received infusion rates equivalent to either the 60 micrograms per kilogram per hour (μg/kg/h) or 90 μg/kg/h group.
  Interventions: Drug: Placebo
- SAGE-547 60 μg/kg/h (Experimental): Participants received a 4-hour titration period of 30 μg/kg/h (0 to 4 hours), then 60 μg/kg/h (4 to 56 hours), followed by a taper to 30 μg/kg/h (56 to 60 hours).
  Interventions: Drug: SAGE-547 60 μg/kg/h
- SAGE-547 90 μg/kg/h (Experimental): Participants received a 4-hour dose titration period of 30 μg/kg/h (0 to 4 hours), then 60 μg/kg/h (4 to 24 hours), then 90 μg/kg/h (24 to 52 hours), followed by a taper to 60 μg/kg/h (52 to 56 hours), and 30 μg/kg/h (56 to 60 hours).
  Interventions: Drug: SAGE-547 90 μg/kg/h

INTERVENTIONS:
Drug: Placebo — Intravenous infusion of matching placebo for either SAGE-547 60 μg/kg/h or 90 μg/kg/h.
  Arms: Placebo
Drug: SAGE-547 60 μg/kg/h — Intravenous infusion of SAGE-547.
  Arms: SAGE-547 60 μg/kg/h
Drug: SAGE-547 90 μg/kg/h — Intravenous infusion of SAGE-547.
  Arms: SAGE-547 90 μg/kg/h

SUMMARY:
The purpose of this study was to determine if SAGE-547 Injection infused intravenously at up to 90 micrograms per kilogram per hour (μg/kg/h) for 60 hours reduces depressive symptoms in participants with severe postpartum depression (PPD) compared to placebo injection as assessed by the change from baseline in Hamilton Rating Scale for Depression (HAM-D) total score.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have ceased lactating at screening; or if still lactating or actively breastfeeding at screening, agreed to temporarily cease giving breastmilk to their infant(s) from just prior to receiving study drug through nine days (Day 12) after the end of the infusion
* Participants had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I)
* Participant had a HAM-D total score of ≥26 at screening and Day 1 (prior to dosing)
* Participant was ≤6 months postpartum at screening
* Participant was amenable to IV therapy

Key Exclusion Criteria:

* Active psychosis
* Attempted suicide associated with index case of postpartum depression
* Medical history of bipolar disorders, schizophrenia, and/or schizoaffective disorder.

Note: Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants with postpartum depression defined as those who a major depressive episode that began no earlier than the third trimester and no later than the first four weeks following delivery, as diagnosed by Structured Clinical Interview Diagnostic and Statistical Manual of Mental Disorders (DSM), 4th Edition Axis I Disorders (SCID-I), a Hamilton Rating Scale for Depression (HAM-D) total score of ≥26 at screening and Day 1 (prior to dosing), and who were ≤6 months postpartum at screening.
Enrollment: 138 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-24 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Sage Therapeutics
Locations (30):
- United States (30):
  - Sage Investigational Site, Chandler, Arizona
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Ventura, California
  - Sage Investigational Site, Gainesville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Miramar, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Pinellas Park, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Hoffman Estates, Illinois
  - Sage Investigational Site, Wichita, Kansas
  - Sage Investigational Site, Edgewood, Kentucky
  - Sage Investigational Site, Owensboro, Kentucky
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Glen Oaks, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Columbus, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, San Antonio, Texas
  - Sage Investigational Site, Orem, Utah

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Derived] Gerbasi ME, Meltzer-Brody S, Acaster S, Fridman M, Bonthapally V, Hodgkins P, Kanes SJ, Eldar-Lissai A. Brexanolone in Postpartum Depression: Post Hoc Analyses to Help Inform Clinical Decision-Making. J Womens Health (Larchmt). 2021 Mar;30(3):385-392. doi: 10.1089/jwh.2020.8483. Epub 2020 Nov 12. PMID 33181049
- [Derived] Meltzer-Brody S, Colquhoun H, Riesenberg R, Epperson CN, Deligiannidis KM, Rubinow DR, Li H, Sankoh AJ, Clemson C, Schacterle A, Jonas J, Kanes S. Brexanolone injection in post-partum depression: two multicentre, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet. 2018 Sep 22;392(10152):1058-1070. doi: 10.1016/S0140-6736(18)31551-4. Epub 2018 Aug 31. Erratum In: Lancet. 2018 Sep 29;392(10153):1116. doi: 10.1016/S0140-6736(18)32288-8. PMID 30177236
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 centers in United States from 01 August 2016 to 19 October 2017.
Pre-assignment Details: A total of 138 participants were randomized into the study to receive either placebo or SAGE-547. Forty-three received placebo, and 79 received SAGE-547.
Period: Overall Study
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Started | 46 | 47 | 45
Participants Who Received Study Drug | 43 | 38 | 41
Completed | 42 | 35 | 36
Not Completed | 4 | 12 | 9
Not completed — Withdrawal by Subject | 0 | 2 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Randomized but not dosed | 3 | 9 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants who started study drug infusion, had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment.
Groups:
- Placebo: Participants received infusion rates equivalent to either the 60 μg/kg/h or 90 μg/kg/h group.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h | Total
Number analyzed (Participants) | 43 | 38 | 41 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.13) | 27.7 (6.46) | 27.5 (6.05) | 27.4 (6.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 41 | 122
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Black or African American | 15 | 12 | 8 | 35
  Native Hawaiian & Other Pacific Islander | 0 | 0 | 1 | 1
  White | 27 | 25 | 29 | 81
  Other | 0 | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latina | 7 | 3 | 7 | 17
  Not Hispanic or Latina | 36 | 35 | 34 | 105
Hamilton Rating Scale for Depression (HAM-D) Total Score [Mean (Standard Deviation); unit: score on a scale] — The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression.
  score on a scale | 28.6 (2.54) | 29.0 (2.70) | 28.4 (2.47) | 28.7 (2.55)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 60 Hours in the 17-Item Hamilton Rating Scale for Depression (HAM-D) Total Score
Description: The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hour 60
Population: All randomized participants who started study drug infusion, had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Overall number of participants analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 37 | 39
score on a scale | -14.04 (1.148) | -19.54 (1.231) | -17.72 (1.193)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Mixed effect model for repeated measures (MMRM) was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0013, MMRM; Least Square (LS) Mean Difference = -5.50, 95% CI 2-sided [-8.80 to -2.20], Standard Error of Mean 1.664
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0252, MMRM; LS mean difference = -3.68, 95% CI 2-sided [-6.90 to -0.47], Standard Error of Mean 1.622

2. Secondary Outcome: Change From Baseline in HAM-D Total Score at Day 30
Description: as for outcome 1
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 42 | 35 | 36
score on a scale | -13.82 (1.324) | -19.45 (1.435) | -17.62 (1.400)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0044, MMRM; LS mean difference = -5.63, 95% CI 2-sided [-9.46 to -1.79], Standard Error of Mean 1.936
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0481, MMRM; LS mean difference = -3.79, 95% CI 2-sided [-7.56 to -0.03], Standard Error of Mean 1.899

3. Secondary Outcome: Change From Baseline in HAM-D Total Score
Description: as for outcome 1
Time Frame: Baseline, Hours 2, 4, 8, 12, 24, 36, 48, 72, and Days 7, 14, and 21
Population: All randomized participants who started study drug infusion, had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
score on a scale
  Change at Hour 2 | -5.04 (0.669) | -4.99 (0.721) | -4.89 (0.707)
  Change at Hour 4 | -6.88 (0.841) | -8.99 (0.902) | -7.18 (0.879)
  Change at Hour 8 | -8.13 (0.928) | -10.18 (0.994) | -8.50 (0.966)
  Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Change at Hour 12 | -9.79 (0.992) | -11.04 (1.069) | -9.07 (1.034)
  Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Change at Hour 24 | -10.71 (1.121) | -15.00 (1.199) | -13.03 (1.157)
  Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Change at Hour 36 | -12.58 (1.114) | -17.69 (1.203) | -13.93 (1.157)
  Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Change at Hour 48 | -13.55 (1.195) | -18.04 (1.282) | -16.89 (1.239)
  Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Change at Hour 72 | -14.67 (1.197) | -19.69 (1.285) | -17.19 (1.243)
  Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Change at Day 7 | -13.34 (1.268) | -17.41 (1.353) | -14.93 (1.315)
  Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Change at Day 14 | -14.64 (1.457) | -17.56 (1.586) | -15.64 (1.521)
  Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Change at Day 21 | -13.23 (1.380) | -18.15 (1.529) | -16.74 (1.451)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9591, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-1.83 to 1.93], Standard Error of Mean 0.951
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8677, MMRM; LS mean difference = 0.15, 95% CI 2-sided [-1.66 to 1.97], Standard Error of Mean 0.917
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0827, MMRM; LS mean difference = -2.11, 95% CI 2-sided [-4.51 to 0.28], Standard Error of Mean 1.208
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.7968, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-2.62 to 2.02], Standard Error of Mean 1.172
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1292, MMRM; LS mean difference = -2.04, 95% CI 2-sided [-4.69 to 0.61], Standard Error of Mean 1.336
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p = 0.7801, MMRM; LS mean difference = -0.36, 95% CI 2-sided [-2.94 to 2.21], Standard Error of Mean 1.299
Statistical Analysis 7: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3840, MMRM; LS mean difference = -1.25, 95% CI 2-sided [-4.10 to 1.59], Standard Error of Mean 1.436
Statistical Analysis 8: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.6097, MMRM; LS mean difference = 0.71, 0.71% CI 2-sided [-2.05 to 3.48], Standard Error of Mean 1.395
Statistical Analysis 9: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0094, MMRM; LS mean difference = -4.28, 95% CI 2-sided [-7.50 to -1.07], Standard Error of Mean 1.622
Statistical Analysis 10: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 9]; Test type: Superiority; p = 0.1440, MMRM; LS mean difference = -2.32, 95% CI 2-sided [-5.45 to 0.80], Standard Error of Mean 1.577
Statistical Analysis 11: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0020, MMRM; LS mean difference = -5.12, 95% CI 2-sided [-8.33 to -1.91], Standard Error of Mean 1.620
Statistical Analysis 12: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 11]; Test type: Superiority; p = 0.3906, MMRM; LS mean difference = -1.36, 95% CI 2-sided [-4.47 to 1.76], Standard Error of Mean 1.572
Statistical Analysis 13: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0110, MMRM; LS mean difference = -4.49, 95% CI 2-sided [-7.93 to -1.05], Standard Error of Mean 1.735
Statistical Analysis 14: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 13]; Test type: Superiority; p = 0.0511, MMRM; LS mean difference = -3.33, 95% CI 2-sided [-6.68 to 0.02], Standard Error of Mean 1.690
Statistical Analysis 15: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at hour 72: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0046, MMRM; LS mean difference = -5.02, 95% CI 2-sided [-8.47 to -1.58], Standard Error of Mean 1.738
Statistical Analysis 16: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 15]; Test type: Superiority; p = 0.1389, MMRM; LS mean difference = -2.53, 95% CI 2-sided [-5.88 to 0.83], Standard Error of Mean 1.694
Statistical Analysis 17: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0288, MMRM; LS mean difference = -4.07, 95% CI 2-sided [-7.71 to -0.43], Standard Error of Mean 1.837
Statistical Analysis 18: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 17]; Test type: Superiority; p = 0.3799, MMRM; LS mean difference = -1.58, 95% CI 2-sided [-5.15 to 1.98], Standard Error of Mean 1.797
Statistical Analysis 19: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1747, MMRM; LS mean difference = -2.92, 95% CI 2-sided [-7.16 to 1.32], Standard Error of Mean 2.139
Statistical Analysis 20: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 19]; Test type: Superiority; p = 0.6310, MMRM; LS mean difference = -1.00, 95% CI 2-sided [-5.13 to 3.12], Standard Error of Mean 2.080
Statistical Analysis 21: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0178, MMRM; LS mean difference = -4.92, 95% CI 2-sided [-8.98 to -0.87], Standard Error of Mean 2.045
Statistical Analysis 22: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 3, analysis 21]; Test type: Superiority; p = 0.0786, MMRM; LS mean difference = -3.51, 95% CI 2-sided [-7.43 to 0.41], Standard Error of Mean 1.976

4. Secondary Outcome: Percentage of Participants With HAM-D Response
Description: The HAM-D response is defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
percentage of participants
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | 55.8 | 86.5 | 74.4
  Day 7: number analyzed (Participants) | 43 | 38 | 40
  Day 7 | 48.8 | 68.4 | 52.5
  Day 30: number analyzed (Participants) | 42 | 35 | 36
  Day 30 | 50.0 | 82.9 | 69.4
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hour 60: Generalized estimating equation (GEE) method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. An exchangeable working correlation structure is assumed for the model parameters estimation; Test type: Superiority; p = 0.0052, GEE method; Odds Ratio (OR) = 5.4, 95% CI 2-sided [1.7 to 17.4]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hour 60: GEE method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. An exchangeable working correlation structure is assumed for the model parameters estimation; Test type: Superiority; p = 0.0493, GEE method; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.0 to 6.9]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Day 7: GEE method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. An exchangeable working correlation structure is assumed for the model parameters estimation; Test type: Superiority; p = 0.0572, GEE method; Odds Ratio (OR) = 2.5, 95% CI 2-sided [1.0 to 6.5]
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.6768, GEE method; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.5 to 3.0]
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Day 30: GEE method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. An exchangeable working correlation structure is assumed for the model parameters estimation; Test type: Superiority; p = 0.0035, GEE method; Odds Ratio (OR) = 5.4, 95% CI 2-sided [1.7 to 16.8]
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0347, GEE method; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.1 to 7.8]

5. Secondary Outcome: Percentage of Participants With HAM-D Remission
Description: The HAM-D remission is defined as having a HAM-D total score of ≤7. The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
percentage of participants
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | 16.3 | 51.4 | 30.8
  Day 7: number analyzed (Participants) | 43 | 38 | 40
  Day 7 | 30.2 | 31.6 | 20.0
  Day 30: number analyzed (Participants) | 42 | 35 | 36
  Day 30 | 31.0 | 48.6 | 38.9
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0011, GEE method; Odds Ratio (OR) = 6.0, 95% CI 2-sided [2.1 to 17.8]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0828, GEE method; Odds Ratio (OR) = 2.6, 95% CI 2-sided [0.9 to 7.6]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.7749, GEE method; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.4 to 3.1]
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.3401, GEE method; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.2 to 1.7]
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.1052, GEE method; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.8 to 6.0]
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.3507, GEE method; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.6 to 4.2]

6. Secondary Outcome: Change From Baseline in HAM-D Bech 6 Subscale
Description: The HAM-D Bech 6 subscale score is calculated as the sum of the following six items: Item # 1 (depressed mood), Item # 2 (feelings of guilt), Item # 7 (work and activities), Item # 8 (retardation), Item # 10 (anxiety psychic), and Item # 13 (general somatic symptoms). Each item is scored in a range of 0 to 2 or 0 to 4, with higher scores indicating a greater degree of depression. The scores were transformed to a 100-point scale with a higher score indicating a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
score on a scale
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | -32.60 (2.962) | -44.67 (3.178) | -38.49 (3.081)
  Day 7: number analyzed (Participants) | 43 | 38 | 40
  Day 7 | -29.43 (3.116) | -38.52 (3.327) | -31.67 (3.236)
  Day 30: number analyzed (Participants) | 42 | 35 | 36
  Day 30 | -30.94 (3.122) | -42.62 (3.385) | -39.20 (3.304)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit as the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables are included in the model. All explanatory variables including pooled center are treated as fixed effects; Test type: Superiority; p = 0.0058, MMRM; LS mean difference = -12.07, 95% CI 2-sided [-20.58 to -3.56], Standard Error of Mean 4.294
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.1622, MMRM; LS mean difference = -5.89, 95% CI 2-sided [-14.19 to 2.41], Standard Error of Mean 4.188
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit as the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables are included in the model. All explanatory variables including pooled center are treated as fixed effects; Test type: Superiority; p = 0.0462, MMRM; LS mean difference = -9.09, 95% CI 2-sided [-18.02 to -0.16], Standard Error of Mean 4.510
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.6124, MMRM; LS mean difference = -2.24, 95% CI 2-sided [-10.97 to 6.49], Standard Error of Mean 4.410
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit as the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables are included in the model. All explanatory variables including pooled center are treated as fixed effects; Test type: Superiority; p = 0.0116, MMRM; LS mean difference = -11.68, 95% CI 2-sided [-20.71 to -2.66], Standard Error of Mean 4.556
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 6, analysis 5]; Test type: Superiority; p = 0.0667, MMRM; LS mean difference = -8.26, 95% CI 2-sided [-17.10 to 0.58], Standard Error of Mean 4.464

7. Secondary Outcome: Change From Baseline in HAM-D Individual Item Scores
Description: The HAM-D comprises individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hour 2, Hour 4, Hour 8, Hour 12, Hour 24, Hour 36, Hour 48, Hour 60, Hour 72 and Days 7, 14, 21 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
score on a scale
  Depressed Mood, Change at Hour 2 | -0.54 (0.133) | -0.54 (0.143) | -0.45 (0.139)
  Depressed Mood, Change at Hour 4 | -0.79 (0.165) | -0.97 (0.176) | -0.79 (0.171)
  Depressed Mood, Change at Hour 8 | -1.02 (0.166) | -1.23 (0.178) | -0.94 (0.172)
  Depressed Mood, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Depressed Mood, Change at Hour 12 | -1.33 (0.170) | -1.50 (0.184) | -1.15 (0.177)
  Depressed Mood, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Depressed Mood, Change at Hour 24 | -1.40 (0.163) | -1.40 (0.175) | -1.47 (0.169)
  Depressed Mood, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Depressed Mood, Change at Hour 36 | -1.47 (0.170) | -2.03 (0.184) | -1.49 (0.176)
  Depressed Mood, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Depressed Mood, Change at Hour 48 | -1.58 (0.173) | -2.07 (0.186) | -1.84 (0.180)
  Depressed Mood, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Depressed Mood, Change at Hour 60 | -1.56 (0.169) | -2.27 (0.181) | -1.92 (0.176)
  Depressed Mood, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Depressed Mood, Change at Hour 72 | -1.75 (0.162) | -2.32 (0.174) | -1.97 (0.169)
  Depressed Mood, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Depressed Mood, Change at Day 7 | -1.49 (0.170) | -1.94 (0.182) | -1.55 (0.177)
  Depressed Mood, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Depressed Mood, Change at Day 14 | -1.53 (0.205) | -2.06 (0.225) | -1.65 (0.213)
  Depressed Mood, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Depressed Mood, Change at Day 21 | -1.48 (0.204) | -1.79 (0.229) | -1.75 (0.214)
  Depressed Mood, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Depressed Mood, Change at Day 30 | -1.53 (0.170) | -2.19 (0.186) | -1.97 (0.183)
  Feelings of Guilt, Change at Hour 2 | -0.46 (0.133) | -0.54 (0.143) | -0.40 (0.138)
  Feelings of Guilt, Change at Hour 4 | -0.70 (0.157) | -1.12 (0.168) | -0.84 (0.162)
  Feelings of Guilt, Change at Hour 8 | -0.84 (0.162) | -1.25 (0.173) | -0.94 (0.168)
  Feelings of Guilt, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Feelings of Guilt, Change at Hour 12 | -1.04 (0.164) | -1.25 (0.178) | -0.76 (0.171)
  Feelings of Guilt, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Feelings of Guilt, Change at Hour 24 | -1.04 (0.162) | -1.50 (0.173) | -1.03 (0.167)
  Feelings of Guilt, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Feelings of Guilt, Change at Hour 36 | -1.23 (0.150) | -1.59 (0.162) | -1.26 (0.156)
  Feelings of Guilt, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Feelings of Guilt, Change at Hour 48 | -1.25 (0.152) | -1.64 (0.163) | -1.60 (0.158)
  Feelings of Guilt, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Feelings of Guilt, Change at Hour 60 | -1.23 (0.149) | -1.68 (0.160) | -1.63 (0.155)
  Feelings of Guilt, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Feelings of Guilt, Change at Hour 72 | -1.42 (0.145) | -1.69 (0.157) | -1.57 (0.152)
  Feelings of Guilt, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Feelings of Guilt, Change at Day 7 | -1.18 (0.152) | -1.38 (0.163) | -1.36 (0.159)
  Feelings of Guilt, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Feelings of Guilt, Change at Day 14 | -1.33 (0.158) | -1.49 (0.173) | -1.56 (0.169)
  Feelings of Guilt, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Feelings of Guilt, Change at Day 21 | -1.10 (0.162) | -1.51 (0.181) | -1.51 (0.171)
  Feelings of Guilt, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Feelings of Guilt, Change at Day 30 | -1.40 (0.149) | -1.61 (0.163) | -1.62 (0.161)
  Suicide, Change at Hour 2 | -0.57 (0.101) | -0.87 (0.107) | -0.48 (0.104)
  Suicide, Change at Hour 4 | -0.64 (0.098) | -0.92 (0.105) | -0.61 (0.101)
  Suicide, Change at Hour 8 | -0.81 (0.088) | -1.00 (0.094) | -0.63 (0.091)
  Suicide, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Suicide, Change at Hour 12 | -0.92 (0.089) | -0.89 (0.096) | -0.66 (0.092)
  Suicide, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Suicide, Change at Hour 24 | -0.87 (0.086) | -0.96 (0.092) | -0.68 (0.088)
  Suicide, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Suicide, Change at Hour 36 | -0.90 (0.068) | -1.00 (0.074) | -0.75 (0.071)
  Suicide, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Suicide, Change at Hour 48 | -0.88 (0.063) | -0.94 (0.069) | -0.95 (0.066)
  Suicide, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Suicide, Change at Hour 60 | -0.81 (0.065) | -1.03 (0.071) | -0.98 (0.069)
  Suicide, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Suicide, Change at Hour 72 | -0.88 (0.068) | -1.01 (0.074) | -0.90 (0.071)
  Suicide, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Suicide, Change at Day 7 | -0.71 (0.089) | -0.90 (0.095) | -0.77 (0.093)
  Suicide, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Suicide, Change at Day 14 | -0.92 (0.084) | -0.99 (0.093) | -0.80 (0.090)
  Suicide, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Suicide, Change at Day 21 | -0.61 (0.133) | -0.80 (0.152) | -0.88 (0.141)
  Suicide, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Suicide, Change at Day 30 | -0.76 (0.080) | -0.99 (0.088) | -0.88 (0.086)
  Insomnia - Early, Change at Hour 2 | -0.27 (0.078) | -0.04 (0.084) | -0.19 (0.082)
  Insomnia - Early, Change at Hour 4 | -0.29 (0.097) | -0.22 (0.104) | -0.29 (0.100)
  Insomnia - Early, Change at Hour 8 | -0.29 (0.103) | -0.17 (0.110) | -0.36 (0.107)
  Insomnia - Early, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Insomnia - Early, Change at Hour 12 | -0.22 (0.092) | -0.25 (0.100) | -0.26 (0.097)
  Insomnia - Early, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Insomnia - Early, Change at Hour 24 | -0.47 (0.138) | -1.10 (0.149) | -0.87 (0.142)
  Insomnia - Early, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Insomnia - Early, Change at Hour 36 | -0.55 (0.142) | -1.16 (0.155) | -0.84 (0.147)
  Insomnia - Early, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Early, Change at Hour 48 | -0.76 (0.144) | -1.07 (0.155) | -1.27 (0.149)
  Insomnia - Early, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Insomnia - Early, Change at Hour 60 | -0.85 (0.140) | -1.10 (0.151) | -1.19 (0.146)
  Insomnia - Early, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Early, Change at Hour 72 | -0.57 (0.142) | -0.96 (0.153) | -0.91 (0.148)
  Insomnia - Early, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Insomnia - Early, Change at Day 7 | -0.69 (0.144) | -1.20 (0.154) | -0.97 (0.150)
  Insomnia - Early, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Insomnia - Early, Change at Day 14 | -0.97 (0.174) | -1.19 (0.192) | -1.06 (0.182)
  Insomnia - Early, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Insomnia - Early, Change at Day 21 | -0.69 (0.154) | -1.28 (0.173) | -1.11 (0.160)
  Insomnia - Early, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Insomnia - Early, Change at Day 30 | -0.67 (0.141) | -1.34 (0.155) | -1.09 (0.153)
  Insomnia - Middle, Change at Hour 2 | -0.13 (0.073) | 0.03 (0.078) | -0.17 (0.076)
  Insomnia - Middle, Change at Hour 4 | -0.16 (0.096) | -0.21 (0.102) | -0.24 (0.099)
  Insomnia - Middle, Change at Hour 8 | -0.20 (0.099) | -0.16 (0.105) | -0.32 (0.102)
  Insomnia - Middle, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Insomnia - Middle, Change at Hour 12 | -0.16 (0.091) | -0.18 (0.098) | -0.22 (0.095)
  Insomnia - Middle, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Insomnia - Middle, Change at Hour 24 | -0.57 (0.135) | -0.98 (0.145) | -0.93 (0.139)
  Insomnia - Middle, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Insomnia - Middle, Change at Hour 36 | -0.74 (0.130) | -1.03 (0.141) | -1.02 (0.135)
  Insomnia - Middle, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Middle, Change at Hour 48 | -0.90 (0.132) | -1.17 (0.142) | -1.19 (0.137)
  Insomnia - Middle, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Insomnia - Middle, Change at Hour 60 | -0.83 (0.130) | -1.22 (0.140) | -1.23 (0.135)
  Insomnia - Middle, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Middle, Change at Hour 72 | -0.93 (0.132) | -1.22 (0.143) | -1.09 (0.138)
  Insomnia - Middle, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Insomnia - Middle, Change at Day 7 | -0.95 (0.128) | -1.05 (0.136) | -0.87 (0.133)
  Insomnia - Middle, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Insomnia - Middle, Change at Day 14 | -0.72 (0.146) | -1.36 (0.161) | -0.98 (0.154)
  Insomnia - Middle, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Insomnia - Middle, Change at Day 21 | -0.77 (0.146) | -1.27 (0.164) | -0.90 (0.152)
  Insomnia - Middle, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Insomnia - Middle, Change at Day 30 | -0.78 (0.134) | -1.21 (0.147) | -0.99 (0.144)
  Insomnia - Late, Change at Hour 2 | -0.16 (0.090) | 0.01 (0.096) | -0.22 (0.094)
  Insomnia - Late, Change at Hour 4 | -0.16 (0.104) | -0.12 (0.111) | -0.34 (0.108)
  Insomnia - Late, Change at Hour 8 | -0.14 (0.103) | -0.20 (0.110) | -0.37 (0.106)
  Insomnia - Late, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Insomnia - Late, Change at Hour 12 | -0.16 (0.103) | -0.01 (0.111) | -0.31 (0.107)
  Insomnia - Late, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Insomnia - Late, Change at Hour 24 | -0.68 (0.123) | -0.94 (0.133) | -0.95 (0.127)
  Insomnia - Late, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Insomnia - Late, Change at Hour 36 | -0.75 (0.127) | -0.91 (0.139) | -0.90 (0.132)
  Insomnia - Late, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Late, Change at Hour 48 | -0.89 (0.125) | -1.16 (0.135) | -1.15 (0.130)
  Insomnia - Late, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Insomnia - Late, Change at Hour 60 | -0.89 (0.121) | -1.16 (0.130) | -1.22 (0.126)
  Insomnia - Late, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Insomnia - Late, Change at Hour 72 | -1.07 (0.121) | -1.13 (0.131) | -1.12 (0.126)
  Insomnia - Late, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Insomnia - Late, Change at Day 7 | -0.89 (0.126) | -0.80 (0.135) | -1.04 (0.132)
  Insomnia - Late, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Insomnia - Late, Change at Day 14 | -0.79 (0.155) | -0.96 (0.172) | -0.86 (0.164)
  Insomnia - Late, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Insomnia - Late, Change at Day 21 | -0.77 (0.157) | -0.89 (0.176) | -0.74 (0.164)
  Insomnia - Late, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Insomnia - Late, Change at Day 30 | -0.77 (0.130) | -1.03 (0.143) | -1.09 (0.140)
  Work and Activities, Change at Hour 2 | -0.30 (0.105) | -0.43 (0.113) | -0.25 (0.111)
  Work and Activities, Change at Hour 4 | -0.51 (0.126) | -0.74 (0.135) | -0.43 (0.131)
  Work and Activities, Change at Hour 8 | -0.81 (0.160) | -0.95 (0.170) | -0.67 (0.165)
  Work and Activities, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Work and Activities, Change at Hour 12 | -1.02 (0.160) | -1.20 (0.173) | -0.83 (0.166)
  Work and Activities, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Work and Activities, Change at Hour 24 | -1.07 (0.169) | -1.19 (0.180) | -1.04 (0.174)
  Work and Activities, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Work and Activities, Change at Hour 36 | -1.39 (0.162) | -1.77 (0.176) | -1.09 (0.168)
  Work and Activities, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Work and Activities, Change at Hour 48 | -1.51 (0.179) | -1.80 (0.192) | -1.57 (0.185)
  Work and Activities, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Work and Activities, Change at Hour 60 | -1.46 (0.171) | -2.04 (0.184) | -1.70 (0.178)
  Work and Activities, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Work and Activities, Change at Hour 72 | -1.67 (0.164) | -2.18 (0.177) | -1.67 (0.171)
  Work and Activities, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Work and Activities, Change at Day 7 | -1.39 (0.176) | -1.82 (0.187) | -1.57 (0.182)
  Work and Activities, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Work and Activities, Change at Day 14 | -1.58 (0.198) | -1.57 (0.218) | -1.60 (0.208)
  Work and Activities, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Work and Activities, Change at Day 21 | -1.35 (0.191) | -1.96 (0.214) | -1.87 (0.200)
  Work and Activities, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Work and Activities, Change at Day 30 | -1.55 (0.174) | -2.08 (0.189) | -1.93 (0.185)
  Retardation, Change at Hour 2 | -0.18 (0.084) | 0.17 (0.090) | -0.01 (0.087)
  Retardation, Change at Hour 4 | -0.34 (0.090) | -0.02 (0.096) | -0.03 (0.093)
  Retardation, Change at Hour 8 | -0.36 (0.092) | -0.20 (0.098) | -0.16 (0.095)
  Retardation, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Retardation, Change at Hour 12 | -0.57 (0.099) | -0.47 (0.107) | -0.42 (0.103)
  Retardation, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Retardation, Change at Hour 24 | -0.48 (0.092) | -0.47 (0.099) | -0.47 (0.095)
  Retardation, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Retardation, Change at Hour 36 | -0.71 (0.103) | -0.87 (0.112) | -0.65 (0.107)
  Retardation, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Retardation, Change at Hour 48 | -0.57 (0.098) | -0.70 (0.105) | -0.60 (0.101)
  Retardation, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Retardation, Change at Hour 60 | -0.76 (0.090) | -0.84 (0.097) | -0.74 (0.094)
  Retardation, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Retardation, Change at Hour 72 | -0.67 (0.092) | -0.87 (0.099) | -0.80 (0.096)
  Retardation, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Retardation, Change at Day 7 | -0.67 (0.091) | -1.02 (0.097) | -0.70 (0.095)
  Retardation, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Retardation, Change at Day 14 | -0.74 (0.117) | -0.87 (0.128) | -0.77 (0.123)
  Retardation, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Retardation, Change at Day 21 | -0.72 (0.104) | -1.05 (0.115) | -0.81 (0.108)
  Retardation, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Retardation, Change at Day 30 | -0.66 (0.088) | -1.08 (0.096) | -0.91 (0.095)
  Agitation, Change at Hour 2 | -0.46 (0.108) | -0.52 (0.115) | -0.45 (0.111)
  Agitation, Change at Hour 4 | -0.56 (0.103) | -0.70 (0.109) | -0.52 (0.106)
  Agitation, Change at Hour 8 | -0.51 (0.112) | -0.68 (0.119) | -0.55 (0.116)
  Agitation, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Agitation, Change at Hour 12 | -0.56 (0.114) | -0.65 (0.123) | -0.59 (0.118)
  Agitation, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Agitation, Change at Hour 24 | -0.54 (0.108) | -0.86 (0.115) | -0.69 (0.110)
  Agitation, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Agitation, Change at Hour 36 | -0.63 (0.111) | -0.82 (0.121) | -0.74 (0.115)
  Agitation, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Agitation, Change at Hour 48 | -0.74 (0.098) | -0.78 (0.105) | -0.78 (0.102)
  Agitation, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Agitation, Change at Hour 60 | -0.58 (0.105) | -0.85 (0.113) | -0.70 (0.110)
  Agitation, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Agitation, Change at Hour 72 | -0.65 (0.112) | -0.85 (0.120) | -0.82 (0.116)
  Agitation, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Agitation, Change at Day 7 | -0.60 (0.098) | -0.78 (0.104) | -0.66 (0.102)
  Agitation, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Agitation, Change at Day 14 | -0.87 (0.114) | -0.75 (0.126) | -0.82 (0.121)
  Agitation, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Agitation, Change at Day 21 | -0.61 (0.142) | -0.69 (0.161) | -0.76 (0.149)
  Agitation, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Agitation, Change at Day 30 | -0.64 (0.112) | -0.80 (0.122) | -0.62 (0.121)
  Anxiety Psychic, Change at Hour 2 | -0.60 (0.134) | -0.70 (0.144) | -0.76 (0.140)
  Anxiety Psychic, Change at Hour 4 | -0.90 (0.158) | -1.26 (0.169) | -1.12 (0.164)
  Anxiety Psychic, Change at Hour 8 | -1.25 (0.161) | -1.41 (0.172) | -1.22 (0.167)
  Anxiety Psychic, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Anxiety Psychic, Change at Hour 12 | -1.39 (0.154) | -1.52 (0.167) | -1.35 (0.161)
  Anxiety Psychic, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Anxiety Psychic, Change at Hour 24 | -1.16 (0.148) | -1.79 (0.159) | -1.59 (0.153)
  Anxiety Psychic, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Anxiety Psychic, Change at Hour 36 | -1.37 (0.149) | -1.99 (0.162) | -1.41 (0.155)
  Anxiety Psychic, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Anxiety Psychic, Change at Hour 48 | -1.41 (0.149) | -1.86 (0.161) | -1.71 (0.156)
  Anxiety Psychic, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Anxiety Psychic, Change at Hour 60 | -1.48 (0.141) | -1.97 (0.152) | -1.64 (0.149)
  Anxiety Psychic, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Anxiety Psychic, Change at Hour 72 | -1.55 (0.152) | -1.84 (0.164) | -1.61 (0.159)
  Anxiety Psychic, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Anxiety Psychic, Change at Day 7 | -1.25 (0.149) | -1.44 (0.160) | -1.30 (0.156)
  Anxiety Psychic, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Anxiety Psychic, Change at Day 14 | -1.42 (0.184) | -1.45 (0.204) | -1.17 (0.195)
  Anxiety Psychic, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Anxiety Psychic, Change at Day 21 | -1.17 (0.197) | -1.26 (0.221) | -1.34 (0.207)
  Anxiety Psychic, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Anxiety Psychic, Change at Day 30 | -1.15 (0.161) | -1.45 (0.176) | -1.43 (0.173)
  Anxiety Somatic, Change at Hour 2 | -0.56 (0.133) | -0.67 (0.142) | -0.75 (0.137)
  Anxiety Somatic, Change at Hour 4 | -0.86 (0.144) | -1.09 (0.154) | -0.88 (0.149)
  Anxiety Somatic, Change at Hour 8 | -0.79 (0.135) | -1.22 (0.145) | -1.05 (0.140)
  Anxiety Somatic, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Anxiety Somatic, Change at Hour 12 | -0.86 (0.130) | -1.16 (0.141) | -0.91 (0.135)
  Anxiety Somatic, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Anxiety Somatic, Change at Hour 24 | -0.77 (0.116) | -1.24 (0.125) | -1.12 (0.120)
  Anxiety Somatic, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Anxiety Somatic, Change at Hour 36 | -0.86 (0.127) | -1.34 (0.140) | -1.08 (0.133)
  Anxiety Somatic, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Anxiety Somatic, Change at Hour 48 | -0.86 (0.125) | -1.42 (0.136) | -1.20 (0.131)
  Anxiety Somatic, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Anxiety Somatic, Change at Hour 60 | -1.00 (0.122) | -1.58 (0.132) | -1.31 (0.128)
  Anxiety Somatic, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Anxiety Somatic, Change at Hour 72 | -0.91 (0.131) | -1.58 (0.142) | -1.29 (0.137)
  Anxiety Somatic, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Anxiety Somatic, Change at Day 7 | -0.91 (0.134) | -1.28 (0.143) | -0.98 (0.140)
  Anxiety Somatic, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Anxiety Somatic, Change at Day 14 | -0.70 (0.153) | -1.08 (0.169) | -0.88 (0.162)
  Anxiety Somatic, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Anxiety Somatic, Change at Day 21 | -0.94 (0.155) | -1.40 (0.175) | -1.05 (0.163)
  Anxiety Somatic, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Anxiety Somatic, Change at Day 30 | -0.80 (0.151) | -1.40 (0.166) | -0.99 (0.163)
  Somatic Symptoms GI, Change at Hour 2 | -0.28 (0.110) | -0.29 (0.118) | -0.30 (0.114)
  Somatic Symptoms GI, Change at Hour 4 | -0.28 (0.103) | -0.55 (0.111) | -0.44 (0.107)
  Somatic Symptoms GI, Change at Hour 8 | -0.42 (0.109) | -0.60 (0.117) | -0.57 (0.113)
  Somatic Symptoms GI, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Somatic Symptoms GI, Change at Hour 12 | -0.51 (0.111) | -0.79 (0.121) | -0.56 (0.116)
  Somatic Symptoms GI, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Somatic Symptoms GI, Change at Hour 24 | -0.47 (0.115) | -0.88 (0.123) | -0.79 (0.118)
  Somatic Symptoms GI, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Somatic Symptoms GI, Change at Hour 36 | -0.54 (0.111) | -1.14 (0.122) | -0.78 (0.116)
  Somatic Symptoms GI, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Somatic Symptoms GI, Change at Hour 48 | -0.61 (0.110) | -1.16 (0.119) | -0.84 (0.115)
  Somatic Symptoms GI, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Somatic Symptoms GI, Change at Hour 60 | -0.82 (0.100) | -1.24 (0.109) | -0.96 (0.106)
  Somatic Symptoms GI, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Somatic Symptoms GI, Change at Hour 72 | -0.68 (0.102) | -1.23 (0.111) | -1.01 (0.107)
  Somatic Symptoms GI, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Somatic Symptoms GI, Change at Day 7 | -0.63 (0.114) | -1.00 (0.123) | -0.66 (0.119)
  Somatic Symptoms GI, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Somatic Symptoms GI, Change at Day 14 | -0.77 (0.126) | -1.03 (0.139) | -0.89 (0.134)
  Somatic Symptoms GI, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Somatic Symptoms GI, Change at Day 21 | -0.70 (0.132) | -1.17 (0.149) | -0.91 (0.139)
  Somatic Symptoms GI, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Somatic Symptoms GI, Change at Day 30 | -0.82 (0.112) | -1.14 (0.123) | -0.91 (0.121)
  Somatic Symptoms General, Change at Hour 2 | -0.23 (0.086) | -0.28 (0.092) | -0.14 (0.089)
  Somatic Symptoms General, Change at Hour 4 | -0.27 (0.093) | -0.44 (0.099) | -0.33 (0.096)
  Somatic Symptoms General, Change at Hour 8 | -0.27 (0.093) | -0.33 (0.099) | -0.28 (0.096)
  Somatic Symptoms General, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Somatic Symptoms General, Change at Hour 12 | -0.51 (0.108) | -0.50 (0.117) | -0.49 (0.113)
  Somatic Symptoms General, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Somatic Symptoms General, Change at Hour 24 | -0.60 (0.119) | -0.67 (0.127) | -0.55 (0.122)
  Somatic Symptoms General, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Somatic Symptoms General, Change at Hour 36 | -0.64 (0.111) | -0.70 (0.122) | -0.79 (0.116)
  Somatic Symptoms General, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Somatic Symptoms General, Change at Hour 48 | -0.67 (0.113) | -1.05 (0.122) | -0.90 (0.117)
  Somatic Symptoms General, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Somatic Symptoms General, Change at Hour 60 | -0.78 (0.111) | -1.06 (0.120) | -0.95 (0.117)
  Somatic Symptoms General, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Somatic Symptoms General, Change at Hour 72 | -0.81 (0.113) | -1.26 (0.121) | -1.00 (0.117)
  Somatic Symptoms General, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Somatic Symptoms General, Change at Day 7 | -0.62 (0.121) | -0.91 (0.129) | -0.61 (0.125)
  Somatic Symptoms General, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Somatic Symptoms General, Change at Day 14 | -0.64 (0.138) | -0.92 (0.152) | -0.59 (0.144)
  Somatic Symptoms General, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Somatic Symptoms General, Change at Day 21 | -0.55 (0.138) | -1.04 (0.154) | -0.72 (0.144)
  Somatic Symptoms General, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Somatic Symptoms General, Change at Day 30 | -0.66 (0.129) | -1.00 (0.140) | -0.95 (0.137)
  Genital Symptoms, Change at Hour 2 | 0.00 (0.055) | 0.00 (0.059) | -0.16 (0.057)
  Genital Symptoms, Change at Hour 4 | 0.00 (0.067) | -0.11 (0.072) | -0.13 (0.069)
  Genital Symptoms, Change at Hour 8 | -0.07 (0.087) | -0.16 (0.093) | -0.16 (0.090)
  Genital Symptoms, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Genital Symptoms, Change at Hour 12 | -0.07 (0.075) | -0.08 (0.082) | -0.24 (0.079)
  Genital Symptoms, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Genital Symptoms, Change at Hour 24 | -0.16 (0.100) | -0.28 (0.106) | -0.28 (0.102)
  Genital Symptoms, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Genital Symptoms, Change at Hour 36 | -0.23 (0.102) | -0.46 (0.111) | -0.51 (0.106)
  Genital Symptoms, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Genital Symptoms, Change at Hour 48 | -0.35 (0.107) | -0.46 (0.115) | -0.63 (0.110)
  Genital Symptoms, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Genital Symptoms, Change at Hour 60 | -0.35 (0.108) | -0.48 (0.116) | -0.67 (0.112)
  Genital Symptoms, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Genital Symptoms, Change at Hour 72 | -0.32 (0.107) | -0.57 (0.115) | -0.72 (0.110)
  Genital Symptoms, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Genital Symptoms, Change at Day 7 | -0.51 (0.113) | -0.71 (0.120) | -0.79 (0.117)
  Genital Symptoms, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Genital Symptoms, Change at Day 14 | -0.49 (0.131) | -0.70 (0.144) | -0.83 (0.138)
  Genital Symptoms, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Genital Symptoms, Change at Day 21 | -0.68 (0.141) | -0.90 (0.159) | -0.87 (0.147)
  Genital Symptoms, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Genital Symptoms, Change at Day 30 | -0.82 (0.131) | -0.97 (0.143) | -0.95 (0.140)
  Hypochondriasis, Change at Hour 2 | -0.23 (0.105) | -0.29 (0.113) | -0.34 (0.109)
  Hypochondriasis, Change at Hour 4 | -0.32 (0.111) | -0.39 (0.119) | -0.34 (0.116)
  Hypochondriasis, Change at Hour 8 | -0.23 (0.114) | -0.47 (0.122) | -0.41 (0.118)
  Hypochondriasis, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Hypochondriasis, Change at Hour 12 | -0.32 (0.109) | -0.41 (0.118) | -0.44 (0.114)
  Hypochondriasis, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Hypochondriasis, Change at Hour 24 | -0.39 (0.105) | -0.55 (0.112) | -0.48 (0.109)
  Hypochondriasis, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Hypochondriasis, Change at Hour 36 | -0.39 (0.104) | -0.61 (0.113) | -0.49 (0.109)
  Hypochondriasis, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Hypochondriasis, Change at Hour 48 | -0.49 (0.105) | -0.63 (0.113) | -0.58 (0.109)
  Hypochondriasis, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hypochondriasis, Change at Hour 60 | -0.49 (0.100) | -0.60 (0.108) | -0.59 (0.105)
  Hypochondriasis, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Hypochondriasis, Change at Hour 72 | -0.60 (0.098) | -0.66 (0.106) | -0.55 (0.103)
  Hypochondriasis, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Hypochondriasis, Change at Day 7 | -0.49 (0.095) | -0.68 (0.102) | -0.58 (0.100)
  Hypochondriasis, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Hypochondriasis, Change at Day 14 | -0.54 (0.120) | -0.59 (0.132) | -0.51 (0.127)
  Hypochondriasis, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Hypochondriasis, Change at Day 21 | -0.84 (0.107) | -0.80 (0.119) | -0.57 (0.114)
  Hypochondriasis, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Hypochondriasis, Change at Day 30 | -0.60 (0.099) | -0.66 (0.109) | -0.60 (0.108)
  Loss of Weight, Change at Hour 2 | -0.05 (0.057) | 0.03 (0.061) | 0.06 (0.059)
  Loss of Weight, Change at Hour 4 | -0.07 (0.052) | -0.04 (0.055) | 0.01 (0.054)
  Loss of Weight, Change at Hour 8 | -0.07 (0.060) | -0.02 (0.064) | -0.04 (0.062)
  Loss of Weight, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Loss of Weight, Change at Hour 12 | -0.09 (0.068) | 0.03 (0.074) | -0.09 (0.071)
  Loss of Weight, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Loss of Weight, Change at Hour 24 | -0.07 (0.084) | -0.12 (0.090) | -0.24 (0.086)
  Loss of Weight, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Loss of Weight, Change at Hour 36 | -0.14 (0.076) | -0.10 (0.082) | -0.19 (0.079)
  Loss of Weight, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Loss of Weight, Change at Hour 48 | -0.05 (0.083) | -0.12 (0.089) | -0.26 (0.086)
  Loss of Weight, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Loss of Weight, Change at Hour 60 | -0.09 (0.095) | -0.26 (0.102) | -0.35 (0.098)
  Loss of Weight, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Loss of Weight, Change at Hour 72 | -0.14 (0.090) | -0.20 (0.097) | -0.26 (0.094)
  Loss of Weight, Change at Day 7: number analyzed (Participants) | 43 | 38 | 39
  Loss of Weight, Change at Day 7 | -0.30 (0.129) | -0.36 (0.137) | -0.60 (0.135)
  Loss of Weight, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Loss of Weight, Change at Day 14 | -0.43 (0.150) | -0.42 (0.164) | -0.64 (0.158)
  Loss of Weight, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Loss of Weight, Change at Day 21 | -0.49 (0.160) | -0.59 (0.177) | -0.61 (0.169)
  Loss of Weight, Change at Day 30: number analyzed (Participants) | 42 | 35 | 35
  Loss of Weight, Change at Day 30 | -0.24 (0.133) | -0.55 (0.144) | -0.48 (0.143)
  Insight, Change at Hour 2 | -0.01 (0.037) | 0.02 (0.040) | 0.02 (0.039)
  Insight, Change at Hour 4 | -0.01 (0.037) | -0.01 (0.040) | 0.04 (0.039)
  Insight, Change at Hour 8 | -0.03 (0.037) | -0.04 (0.040) | 0.04 (0.039)
  Insight, Change at Hour 12: number analyzed (Participants) | 43 | 36 | 40
  Insight, Change at Hour 12 | -0.03 (0.037) | -0.06 (0.041) | 0.07 (0.039)
  Insight, Change at Hour 24: number analyzed (Participants) | 42 | 37 | 41
  Insight, Change at Hour 24 | 0.04 (0.038) | -0.01 (0.040) | 0.04 (0.039)
  Insight, Change at Hour 36: number analyzed (Participants) | 43 | 35 | 40
  Insight, Change at Hour 36 | -0.03 (0.037) | -0.04 (0.041) | -0.01 (0.039)
  Insight, Change at Hour 48: number analyzed (Participants) | 43 | 37 | 40
  Insight, Change at Hour 48 | -0.03 (0.037) | 0.02 (0.040) | 0.02 (0.039)
  Insight, Change at Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Insight, Change at Hour 60 | -0.06 (0.037) | -0.06 (0.040) | -0.09 (0.039)
  Insight, Change at Hour 72: number analyzed (Participants) | 43 | 37 | 40
  Insight, Change at Hour 72 | -0.06 (0.037) | -0.01 (0.040) | -0.06 (0.039)
  Insight, Change at Day 7: number analyzed (Participants) | 43 | 38 | 40
  Insight, Change at Day 7 | -0.06 (0.037) | -0.06 (0.040) | -0.03 (0.039)
  Insight, Change at Day 14: number analyzed (Participants) | 29 | 23 | 26
  Insight, Change at Day 14 | -0.03 (0.041) | -0.07 (0.045) | -0.09 (0.044)
  Insight, Change at Day 21: number analyzed (Participants) | 29 | 22 | 27
  Insight, Change at Day 21 | -0.10 (0.042) | -0.08 (0.047) | -0.09 (0.044)
  Insight, Change at Day 30: number analyzed (Participants) | 42 | 35 | 36
  Insight, Change at Day 30 | -0.01 (0.038) | -0.06 (0.041) | -0.08 (0.041)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9681, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.39 to 0.37], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.6337, MMRM; LS mean difference = 0.09, 95% CI 2-sided [-0.28 to 0.46], Standard Error of Mean 0.185
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4690, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.64 to 0.30], Standard Error of Mean 0.238
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 3]; Test type: Superiority; p = 0.9905, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.46 to 0.46], Standard Error of Mean 0.232
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3984, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.68 to 0.27], Standard Error of Mean 0.240
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 5]; Test type: Superiority; p = 0.7042, MMRM; LS mean difference = 0.09, 95% CI 2-sided [-0.37 to 0.55], Standard Error of Mean 0.234
Statistical Analysis 7: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4941, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.66 to 0.32], Standard Error of Mean 0.247
Statistical Analysis 8: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 7]; Test type: Superiority; p = 0.4572, MMRM; LS mean difference = 0.18, 95% CI 2-sided [-0.30 to 0.65], Standard Error of Mean 0.240
Statistical Analysis 9: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9866, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.47 to 0.46], Standard Error of Mean 0.236
Statistical Analysis 10: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 9]; Test type: Superiority; p = 0.7490, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.53 to 0.38], Standard Error of Mean 0.229
Statistical Analysis 11: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0235, MMRM; LS mean difference = -0.57, 95% CI 2-sided [-1.06 to -0.08], Standard Error of Mean 0.247
Statistical Analysis 12: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Change Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9286, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.50 to 0.45], Standard Error of Mean 0.239
Statistical Analysis 13: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0544, MMRM; LS mean difference = -0.49, 95% CI 2-sided [-0.99 to 0.01], Standard Error of Mean 0.251
Statistical Analysis 14: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 13]; Test type: Superiority; p = 0.2903, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.74 to 0.22], Standard Error of Mean 0.244
Statistical Analysis 15: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0044, MMRM; LS mean difference = -0.71, 95% CI 2-sided [-1.19 to -0.23], Standard Error of Mean 0.244
Statistical Analysis 16: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 15]; Test type: Superiority; p = 0.1339, MMRM; LS mean difference = -0.36, 95% CI 2-sided [-0.83 to 0.11], Standard Error of Mean 0.238
Statistical Analysis 17: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0149, MMRM; LS mean difference = -0.58, 95% CI 2-sided [-1.04 to -0.11], Standard Error of Mean 0.234
Statistical Analysis 18: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 17]; Test type: Superiority; p = 0.3213, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.68 to 0.22], Standard Error of Mean 0.228
Statistical Analysis 19: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0703, MMRM; LS mean difference = -0.45, 95% CI 2-sided [-0.94 to 0.04], Standard Error of Mean 0.246
Statistical Analysis 20: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 19]; Test type: Superiority; p = 0.8152, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.53 to 0.42], Standard Error of Mean 0.240
Statistical Analysis 21: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0805, MMRM; LS mean difference = -0.53, 95% CI 2-sided [-1.13 to 0.07], Standard Error of Mean 0.301
Statistical Analysis 22: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 21]; Test type: Superiority; p = 0.6964, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.69 to 0.46], Standard Error of Mean 0.291
Statistical Analysis 23: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2998, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.92 to 0.29], Standard Error of Mean 0.304
Statistical Analysis 24: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 23]; Test type: Superiority; p = 0.3448, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.85 to 0.30], Standard Error of Mean 0.291
Statistical Analysis 25: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Depressed Mood, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0089, MMRM; LS mean difference = -0.66, 95% CI 2-sided [-1.15 to -0.17], Standard Error of Mean 0.248
Statistical Analysis 26: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 25]; Test type: Superiority; p = 0.0772, MMRM; LS mean difference = -0.44, 95% CI 2-sided [-0.92 to 0.05], Standard Error of Mean 0.244
Statistical Analysis 27: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6809, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.46 to 0.30], Standard Error of Mean 0.191
Statistical Analysis 28: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 27]; Test type: Superiority; p = 0.7297, MMRM; LS mean difference = 0.06, 95% CI 2-sided [-0.30 to 0.43], Standard Error of Mean 0.185
Statistical Analysis 29: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0626, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.87 to 0.02], Standard Error of Mean 0.226
Statistical Analysis 30: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 29]; Test type: Superiority; p = 0.5196, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.58 to 0.29], Standard Error of Mean 0.220
Statistical Analysis 31: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0772, MMRM; LS mean difference = -0.42, 95% CI 2-sided [-0.88 to 0.05], Standard Error of Mean 0.234
Statistical Analysis 32: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 31]; Test type: Superiority; p = 0.6610, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.55 to 0.35], Standard Error of Mean 0.228
Statistical Analysis 33: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4007, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.67 to 0.27], Standard Error of Mean 0.239
Statistical Analysis 34: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 33]; Test type: Superiority; p = 0.2292, MMRM; LS mean difference = 0.28, 95% CI 2-sided [-0.18 to 0.74], Standard Error of Mean 0.232
Statistical Analysis 35: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0540, MMRM; LS mean difference = -0.45, 95% CI 2-sided [-0.92 to 0.01], Standard Error of Mean 0.234
Statistical Analysis 36: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 35]; Test type: Superiority; p = 0.9590, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.44 to 0.46], Standard Error of Mean 0.227
Statistical Analysis 37: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1048, MMRM; LS mean difference = -0.36, 95% CI 2-sided [-0.79 to 0.08], Standard Error of Mean 0.218
Statistical Analysis 38: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 37]; Test type: Superiority; p = 0.8979, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.44 to 0.39], Standard Error of Mean 0.210
Statistical Analysis 39: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0819, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-0.82 to 0.05], Standard Error of Mean 0.219
Statistical Analysis 40: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 39]; Test type: Superiority; p = 0.1099, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.77 to 0.08], Standard Error of Mean 0.213
Statistical Analysis 41: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0373, MMRM; LS mean difference = -0.45, 95% CI 2-sided [-0.88 to -0.03], Standard Error of Mean 0.215
Statistical Analysis 42: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 41]; Test type: Superiority; p = 0.0577, MMRM; LS mean difference = -0.40, 95% CI 2-sided [-0.81 to 0.01], Standard Error of Mean 0.209
Statistical Analysis 43: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2023, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.69 to 0.15], Standard Error of Mean 0.210
Statistical Analysis 44: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 43]; Test type: Superiority; p = 0.4444, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.56 to 0.25], Standard Error of Mean 0.204
Statistical Analysis 45: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3645, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.64 to 0.24], Standard Error of Mean 0.220
Statistical Analysis 46: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 45]; Test type: Superiority; p = 0.4035, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.60 to 0.24], Standard Error of Mean 0.214
Statistical Analysis 47: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4877, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.62 to 0.30], Standard Error of Mean 0.232
Statistical Analysis 48: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 47]; Test type: Superiority; p = 0.3134, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.68 to 0.22], Standard Error of Mean 0.226
Statistical Analysis 49: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0922, MMRM; LS mean difference = -0.41, 95% CI 2-sided [-0.89 to 0.07], Standard Error of Mean 0.240
Statistical Analysis 50: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 49]; Test type: Superiority; p = 0.0761, MMRM; LS mean difference = -0.41, 95% CI 2-sided [-0.87 to 0.04], Standard Error of Mean 0.230
Statistical Analysis 51: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Feelings of Guilt, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3275, MMRM; LS mean difference = -0.21, 95% CI 2-sided [-0.64 to 0.22], Standard Error of Mean 0.217
Statistical Analysis 52: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 51]; Test type: Superiority; p = 0.3041, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.64 to 0.20], Standard Error of Mean 0.213
Statistical Analysis 53: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0450, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.59 to -0.01], Standard Error of Mean 0.146
Statistical Analysis 54: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 53]; Test type: Superiority; p = 0.5351, MMRM; LS mean difference = 0.09, 95% CI 2-sided [-0.19 to 0.37], Standard Error of Mean 0.143
Statistical Analysis 55: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0525, MMRM; LS men difference = -0.28, 95% CI 2-sided [-0.56 to 0.00], Standard Error of Mean 0.142
Statistical Analysis 56: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 55]; Test type: Superiority; p = 0.7932, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.24 to 0.31], Standard Error of Mean 0.139
Statistical Analysis 57: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1300, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.45 to 0.06], Standard Error of Mean 0.128
Statistical Analysis 58: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 57]; Test type: Superiority; p = 0.1631, MMRM; LS mean difference = 0.17, 95% CI 2-sided [-0.07 to 0.42], Standard Error of Mean 0.125
Statistical Analysis 59: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8215, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.23 to 0.29], Standard Error of Mean 0.129
Statistical Analysis 60: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 59]; Test type: Superiority; p = 0.0380, MMRM; LS mean difference = 0.26, 95% CI 2-sided [0.01 to 0.51], Standard Error of Mean 0.126
Statistical Analysis 61: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5070, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.33 to 0.16], Standard Error of Mean 0.124
Statistical Analysis 62: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 61]; Test type: Superiority; p = 0.1094, MMRM; LS mean difference = 0.19, 95% CI 2-sided [-0.04 to 0.43], Standard Error of Mean 0.120
Statistical Analysis 63: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3112, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.30 to 0.10], Standard Error of Mean 0.099
Statistical Analysis 64: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 63]; Test type: Superiority; p = 0.1345, MMRM; LS mean difference = 0.14, 95% CI 2-sided [-0.05 to 0.33], Standard Error of Mean 0.096
Statistical Analysis 65: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5148, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.24 to 0.12], Standard Error of Mean 0.091
Statistical Analysis 66: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 65]; Test type: Superiority; p = 0.3863, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.25 to 0.10], Standard Error of Mean 0.088
Statistical Analysis 67: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0209, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.41 to -0.03], Standard Error of Mean 0.094
Statistical Analysis 68: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 67]; Test type: Superiority; p = 0.0616, MMRM; LS men difference = -0.17, 95% CI 2-sided [-0.35 to 0.01], Standard Error of Mean 0.092
Statistical Analysis 69: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1860, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.33 to 0.06], Standard Error of Mean 0.099
Statistical Analysis 70: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 69]; Test type: Superiority; p = 0.7730, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.22 to 0.16], Standard Error of Mean 0.095
Statistical Analysis 71: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1593, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.44 to 0.07], Standard Error of Mean 0.129
Statistical Analysis 72: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 71]; Test type: Superiority; p = 0.6371, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.31 to 0.19], Standard Error of Mean 0.126
Statistical Analysis 73: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5655, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.32 to 0.18], Standard Error of Mean 0.124
Statistical Analysis 74: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 73]; Test type: Superiority; p = 0.3326, MMRM; LS mean difference = 0.12, 95% CI 2-sided [-0.12 to 0.36], Standard Error of Mean 0.121
Statistical Analysis 75: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3577, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.59 to 0.22], Standard Error of Mean 0.201
Statistical Analysis 76: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 75]; Test type: Superiority; p = 0.1646, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.66 to 0.11], Standard Error of Mean 0.192
Statistical Analysis 77: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Suicide, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0545, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.46 to 0.00], Standard Error of Mean 0.118
Statistical Analysis 78: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 77]; Test type: Superiority; p = 0.2903, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.35 to 0.11], Standard Error of Mean 0.115
Statistical Analysis 79: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0395, MMRM; LS mean difference = 0.23, 95% CI 2-sided [0.01 to 0.45], Standard Error of Mean 0.112
Statistical Analysis 80: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 79]; Test type: Superiority; p = 0.4690, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.14 to 0.29], Standard Error of Mean 0.108
Statistical Analysis 81: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6066, MMRM; LS difference = 0.07, 95% CI 2-sided [-0.20 to 0.35], Standard Error of Mean 0.139
Statistical Analysis 82: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 81]; Test type: Superiority; p = 0.9737, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.26 to 0.27], Standard Error of Mean 0.136
Statistical Analysis 83: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4030, MMRM; LS mean difference = 0.12, 95% CI 2-sided [-0.17 to 0.42], Standard Error of Mean 0.148
Statistical Analysis 84: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 83]; Test type: Superiority; p = 0.6357, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.36 to 0.22], Standard Error of Mean 0.145
Statistical Analysis 85: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8605, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.29 to 0.24], Standard Error of Mean 0.134
Statistical Analysis 86: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 85]; Test type: Superiority; p = 0.7534, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.30 to 0.22], Standard Error of Mean 0.130
Statistical Analysis 87: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0021, MMRM; LS mean difference = -0.63, 95% CI 2-sided [-1.03 to -0.23], Standard Error of Mean 0.201
Statistical Analysis 88: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 87]; Test type: Superiority; p = 0.0394, MMRM; LS mean difference = -0.41, 95% CI 2-sided [-0.80 to -0.02], Standard Error of Mean 0.196
Statistical Analysis 89: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0039, Wilcoxon (Mann-Whitney); LS mean difference = -0.61, 95% CI 2-sided [-1.03 to -0.20], Standard Error of Mean 0.208
Statistical Analysis 90: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 89]; Test type: Superiority; p = 0.1591, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.69 to 0.11], Standard Error of Mean 0.202
Statistical Analysis 91: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1402, MMRM; LS mean difference = -0.31, 95% CI 2-sided [-0.73 to 0.10], Standard Error of Mean 0.210
Statistical Analysis 92: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 91]; Test type: Superiority; p = 0.0143, MMRM; LS mean difference = -0.51, 95% CI 2-sided [-0.91 to -0.10], Standard Error of Mean 0.205
Statistical Analysis 93: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2293, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.65 to 0.16], Standard Error of Mean 0.204
Statistical Analysis 94: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 93]; Test type: Superiority; p = 0.0884, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.74 to 0.05], Standard Error of Mean 0.200
Statistical Analysis 95: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0622, MMRM; LS mean difference = -0.39, 95% CI 2-sided [-0.80 to 0.02], Standard Error of Mean 0.207
Statistical Analysis 96: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 95]; Test type: Superiority; p = 0.0955, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.74 to 0.06], Standard Error of Mean 0.202
Statistical Analysis 97: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0173, MMRM; LS mean difference = -0.51, 95% CI 2-sided [-0.92 to -0.09], Standard Error of Mean 0.210
Statistical Analysis 98: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 97]; Test type: Superiority; p = 0.1687, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.69 to 0.12], Standard Error of Mean 0.206
Statistical Analysis 99: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3861, Wilcoxon (Mann-Whitney); LS mean difference = -0.22, 95% CI 2-sided [-0.74 to 0.29], Standard Error of Mean 0.258
Statistical Analysis 100: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 99]; Test type: Superiority; p = 0.7060, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.59 to 0.40], Standard Error of Mean 0.249
Statistical Analysis 101: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0112, MMRM; LS mean difference = -0.59, 95% CI 2-sided [-1.05 to -0.14], Standard Error of Mean 0.230
Statistical Analysis 102: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 101]; Test type: Superiority; p = 0.0570, MMRM; LS mean difference = -0.42, 95% CI 2-sided [-0.86 to 0.01], Standard Error of Mean 0.219
Statistical Analysis 103: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Early, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0018, MMRM; LS mean difference = -0.67, 95% CI 2-sided [-1.08 to -0.26], Standard Error of Mean 0.208
Statistical Analysis 104: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 103]; Test type: Superiority; p = 0.0443, MMRM; LS mean difference = -0.42, 95% CI 2-sided [-0.83 to -0.01], Standard Error of Mean 0.205
Statistical Analysis 105: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1197, MMRM; LS mean difference = 0.16, 95% CI 2-sided [-0.04 to 0.37], Standard Error of Mean 0.104
Statistical Analysis 106: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 105]; Test type: Superiority; p = 0.7171, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.24 to 0.16], Standard Error of Mean 0.101
Statistical Analysis 107: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7151, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.32 to 0.22], Standard Error of Mean 0.138
Statistical Analysis 108: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 107]; Test type: Superiority; p = 0.5210, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.35 to 0.18], Standard Error of Mean 0.134
Statistical Analysis 109: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7332, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.23 to 0.33], Standard Error of Mean 0.142
Statistical Analysis 110: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 109]; Test type: Superiority; p = 0.4163, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.39 to 0.16], Standard Error of Mean 0.139
Statistical Analysis 111: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8625, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.28 to 0.24], Standard Error of Mean 0.132
Statistical Analysis 112: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 111]; Test type: Superiority; p = 0.6196, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.32 to 0.19], Standard Error of Mean 0.128
Statistical Analysis 113: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0373, MMRM; LS mean difference = -0.41, 95% CI 2-sided [-0.80 to -0.02], Standard Error of Mean 0.197
Statistical Analysis 114: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 113]; Test type: Superiority; p = 0.0644, MMRM; LS mean difference = -0.36, 95% CI 2-sided [-0.74 to 0.02], Standard Error of Mean 0.191
Statistical Analysis 115: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1347, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.66 to 0.09], Standard Error of Mean 0.191
Statistical Analysis 116: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 115]; Test type: Superiority; p = 0.1269, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.65 to 0.08], Standard Error of Mean 0.185
Statistical Analysis 117: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1650, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.65 to 0.11], Standard Error of Mean 0.192
Statistical Analysis 118: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 117]; Test type: Superiority; p = 0.1291, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.66 to 0.08], Standard Error of Mean 0.188
Statistical Analysis 119: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0402, MMRM; LS mean difference = -0.39, 95% CI 2-sided [-0.77 to -0.02], Standard Error of Mean 0.189
Statistical Analysis 120: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 119]; Test type: Superiority; p = 0.0342, MMRM; LS mean difference = -0.40, 95% CI 2-sided [-0.76 to -0.03], Standard Error of Mean 0.185
Statistical Analysis 121: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1269, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.68 to 0.09], Standard Error of Mean 0.193
Statistical Analysis 122: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 121]; Test type: Superiority; p = 0.3945, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.53 to 0.21], Standard Error of Mean 0.188
Statistical Analysis 123: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5828, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.47 to 0.26], Standard Error of Mean 0.185
Statistical Analysis 124: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 123]; Test type: Superiority; p = 0.6625, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.28 to 0.44], Standard Error of Mean 0.182
Statistical Analysis 125: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0041, MMRM; LS mean difference = -0.64, 95% CI 2-sided [-1.07 to -0.21], Standard Error of Mean 0.216
Statistical Analysis 126: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 125]; Test type: Superiority; p = 0.2222, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.67 to 0.16], Standard Error of Mean 0.210
Statistical Analysis 127: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0245, MMRM; LS mean difference = -0.50, 95% CI 2-sided [-0.93 to -0.07], Standard Error of Mean 0.218
Statistical Analysis 128: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 127]; Test type: Superiority; p = 0.5119, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.55 to 0.28], Standard Error of Mean 0.209
Statistical Analysis 129: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Middle, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0299, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.82 to -0.04], Standard Error of Mean 0.197
Statistical Analysis 130: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 129]; Test type: Superiority; p = 0.2824, MMRM; LS mean difference = -0.21, 95% CI 2-sided [-0.60 to 0.18], Standard Error of Mean 0.195
Statistical Analysis 131: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1768, MMRM; LS mean difference = 0.18, 95% CI 2-sided [-0.08 to 0.43], Standard Error of Mean 0.129
Statistical Analysis 132: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 131]; Test type: Superiority; p = 0.6498, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.31 to 0.19], Standard Error of Mean 0.126
Statistical Analysis 133: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7689, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.25 to 0.34], Standard Error of Mean 0.150
Statistical Analysis 134: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 133]; Test type: Superiority; p = 0.2236, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.47 to 0.11], Standard Error of Mean 0.146
Statistical Analysis 135: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6952, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.35 to 0.23], Standard Error of Mean 0.148
Statistical Analysis 136: Comparison: Placebo; [analysis description as in outcome 7, analysis 135]; Test type: Superiority; p = 0.1184, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.51 to 0.06], Standard Error of Mean 0.144
Statistical Analysis 137: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3031, MMRM; LS mean difference = 0.15, 95% CI 2-sided [-0.14 to 0.45], Standard Error of Mean 0.149
Statistical Analysis 138: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 137]; Test type: Superiority; p = 0.3091, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.44 to 0.14], Standard Error of Mean 0.145
Statistical Analysis 139: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1525, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.61 to 0.10], Standard Error of Mean 0.179
Statistical Analysis 140: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 139]; Test type: Superiority; p = 0.1214, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.62 to 0.07], Standard Error of Mean 0.174
Statistical Analysis 141: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3811, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.53 to 0.21], Standard Error of Mean 0.187
Statistical Analysis 142: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 141]; Test type: Superiority; p = 0.3851, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.51 to 0.20], Standard Error of Mean 0.180
Statistical Analysis 143: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1373, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.63 to 0.09], Standard Error of Mean 0.182
Statistical Analysis 144: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 143]; Test type: Superiority; p = 0.1360, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.62 to 0.09], Standard Error of Mean 0.177
Statistical Analysis 145: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1264, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.62 to 0.08], Standard Error of Mean 0.176
Statistical Analysis 146: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 145]; Test type: Superiority; p = 0.0567, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.67 to 0.01], Standard Error of Mean 0.172
Statistical Analysis 147: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7447, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.41 to 0.29], Standard Error of Mean 0.176
Statistical Analysis 148: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 147]; Test type: Superiority; p = 0.7727, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.39 to 0.29], Standard Error of Mean 0.172
Statistical Analysis 149: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6590, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.28 to 0.44], Standard Error of Mean 0.183
Statistical Analysis 150: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 149]; Test type: Superiority; p = 0.3951, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.51 to 0.20], Standard Error of Mean 0.180
Statistical Analysis 151: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4576, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.63 to 0.28], Standard Error of Mean 0.230
Statistical Analysis 152: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 151]; Test type: Superiority; p = 0.7609, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.51 to 0.37], Standard Error of Mean 0.223
Statistical Analysis 153: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6220, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.58 to 0.35], Standard Error of Mean 0.234
Statistical Analysis 154: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 153]; Test type: Superiority; p = 0.9081, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.42 to 0.47], Standard Error of Mean 0.225
Statistical Analysis 155: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insomnia - Late, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1668, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.65 to 0.11], Standard Error of Mean 0.191
Statistical Analysis 156: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 155]; Test type: Superiority; p = 0.0935, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.69 to 0.05], Standard Error of Mean 0.189
Statistical Analysis 157: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4038, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.42 to 0.17], Standard Error of Mean 0.150
Statistical Analysis 158: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 157]; Test type: Superiority; p = 0.7559, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.24 to 0.33], Standard Error of Mean 0.145
Statistical Analysis 159: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2006, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.59 to 0.13], Standard Error of Mean 0.181
Statistical Analysis 160: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 159]; Test type: Superiority; p = 0.6334, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.26 to 0.43], Standard Error of Mean 0.175
Statistical Analysis 161: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5431, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.60 to 0.32], Standard Error of Mean 0.230
Statistical Analysis 162: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 161]; Test type: Superiority; p = 0.5278, MMRM; LS mean difference = 0.14, 95% CI 2-sided [-0.30 to 0.59], Standard Error of Mean 0.225
Statistical Analysis 163: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4312, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.64 to 0.28], Standard Error of Mean 0.232
Statistical Analysis 164: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 163]; Test type: Superiority; p = 0.3947, MMRM; LS mean difference = 0.19, 95% CI 2-sided [-0.25 to 0.64], Standard Error of Mean 0.225
Statistical Analysis 165: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6081, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.61 to 0.36], Standard Error of Mean 0.244
Statistical Analysis 166: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 165]; Test type: Superiority; p = 0.8949, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.44 to 0.50], Standard Error of Mean 0.238
Statistical Analysis 167: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1120, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-0.84 to 0.09], Standard Error of Mean 0.236
Statistical Analysis 168: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 167]; Test type: Superiority; p = 0.1842, MMRM; LS mean difference = 0.30, 95% CI 2-sided [-0.15 to 0.76], Standard Error of Mean 0.228
Statistical Analysis 169: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2646, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.81 to 0.22], Standard Error of Mean 0.260
Statistical Analysis 170: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 169]; Test type: Superiority; p = 0.8101, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.56 to 0.44], Standard Error of Mean 0.253
Statistical Analysis 171: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0215, MMRM; LS mean difference = -0.58, 95% CI 2-sided [-1.07 to -0.09], Standard Error of Mean 0.248
Statistical Analysis 172: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 171]; Test type: Superiority; p = 0.3226, MMRM; LS mean difference = -0.24, 95% CI 2-sided [-0.72 to 0.24], Standard Error of Mean 0.242
Statistical Analysis 173: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0339, MMRM; LS mean difference = -0.51, 95% CI 2-sided [-0.98 to -0.04], Standard Error of Mean 0.238
Statistical Analysis 174: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 173]; Test type: Superiority; p = 0.9824, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.46 to 0.47], Standard Error of Mean 0.232
Statistical Analysis 175: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0950, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.93 to 0.08], Standard Error of Mean 0.254
Statistical Analysis 176: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 175]; Test type: Superiority; p = 0.4865, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.67 to 0.32], Standard Error of Mean 0.249
Statistical Analysis 177: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9861, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.57 to 0.58], Standard Error of Mean 0.292
Statistical Analysis 178: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 177]; Test type: Superiority; p = 0.9266, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.59 to 0.54], Standard Error of Mean 0.283
Statistical Analysis 179: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0360, MMRM; LS mean difference = -0.61, 95% CI 2-sided [-1.17 to -0.04], Standard Error of Mean 0.285
Statistical Analysis 180: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 179]; Test type: Superiority; p = 0.0583, MMRM; LS mean difference = -0.52, 95% CI 2-sided [-1.06 to 0.02], Standard Error of Mean 0.273
Statistical Analysis 181: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Work and Activities, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0404, MMRM; LS mean difference = -0.53, 95% CI 2-sided [-1.03 to -0.02], Standard Error of Mean 0.254
Statistical Analysis 182: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 181]; Test type: Superiority; p = 0.1352, MMRM; LS mean difference = -0.37, 95% CI 2-sided [-0.87 to 0.12], Standard Error of Mean 0.249
Statistical Analysis 183: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0056, MMRM; LS mean difference = 0.34, 95% CI 2-sided [0.10 to 0.58], Standard Error of Mean 0.121
Statistical Analysis 184: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 183]; Test type: Superiority; p = 0.1537, MMRM; LS mean difference = 0.17, 95% CI 2-sided [-0.06 to 0.40], Standard Error of Mean 0.118
Statistical Analysis 185: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0142, MMRM; LS mean difference = 0.32, 95% CI 2-sided [0.07 to 0.58], Standard Error of Mean 0.129
Statistical Analysis 186: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 185]; Test type: Superiority; p = 0.0159, MMRM; LS mean difference = 0.31, 95% CI 2-sided [0.06 to 0.56], Standard Error of Mean 0.126
Statistical Analysis 187: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2255, MMRM; LS mean difference = 0.16, 95% CI 2-sided [-0.10 to 0.42], Standard Error of Mean 0.132
Statistical Analysis 188: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 187]; Test type: Superiority; p = 0.1069, MMRM; LS mean difference = 0.21, 95% CI 2-sided [-0.05 to 0.46], Standard Error of Mean 0.129
Statistical Analysis 189: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4932, MMRM; LS mean difference = 0.10, 95% CI 2-sided [-0.19 to 0.39], Standard Error of Mean 0.144
Statistical Analysis 190: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 189]; Test type: Superiority; p = 0.2634, MMRM; LS mean difference = 0.16, 95% CI 2-sided [-0.12 to 0.43], Standard Error of Mean 0.140
Statistical Analysis 191: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9284, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.25 to 0.28], Standard Error of Mean 0.133
Statistical Analysis 192: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 191]; Test type: Superiority; p = 0.9459, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.25 to 0.26], Standard Error of Mean 0.129
Statistical Analysis 193: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2908, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.46 to 0.14], Standard Error of Mean 0.151
Statistical Analysis 194: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 193]; Test type: Superiority; p = 0.6834, MMRM; LS mean difference = 0.06, 95% CI 2-sided [-0.23 to 0.35], Standard Error of Mean 0.146
Statistical Analysis 195: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3579, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.41 to 0.15], Standard Error of Mean 0.142
Statistical Analysis 196: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 195]; Test type: Superiority; p = 0.8270, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.30 to 0.24], Standard Error of Mean 0.138
Statistical Analysis 197: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5292, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.34 to 0.18], Standard Error of Mean 0.130
Statistical Analysis 198: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 197]; Test type: Superiority; p = 0.8790, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.23 to 0.27], Standard Error of Mean 0.127
Statistical Analysis 199: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1347, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.46 to 0.06], Standard Error of Mean 0.133
Statistical Analysis 200: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 199]; Test type: Superiority; p = 0.2874, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.40 to 0.12], Standard Error of Mean 0.129
Statistical Analysis 201: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0086, MMRM; LS mean difference = -0.35, 95% CI 2-sided [-0.61 to -0.09], Standard Error of Mean 0.132
Statistical Analysis 202: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 201]; Test type: Superiority; p = 0.7864, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.29 to 0.22], Standard Error of Mean 0.129
Statistical Analysis 203: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4383, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.48 to 0.21], Standard Error of Mean 0.172
Statistical Analysis 204: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 203]; Test type: Superiority; p = 0.8767, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.36 to 0.31], Standard Error of Mean 0.167
Statistical Analysis 205: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0341, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.63 to -0.03], Standard Error of Mean 0.153
Statistical Analysis 206: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 205]; Test type: Superiority; p = 0.5629, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.38 to 0.21], Standard Error of Mean 0.147
Statistical Analysis 207: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Retardation, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0016, MMRM; LS mean difference = -0.42, 95% CI 2-sided [-0.67 to -0.16], Standard Error of Mean 0.129
Statistical Analysis 208: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 207]; Test type: Superiority; p = 0.0495, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.50 to 0.00], Standard Error of Mean 0.126
Statistical Analysis 209: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7177, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.36 to 0.25], Standard Error of Mean 0.155
Statistical Analysis 210: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 209]; Test type: Superiority; p = 0.9401, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.29 to 0.31], Standard Error of Mean 0.151
Statistical Analysis 211: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3201, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.44 to 0.15], Standard Error of Mean 0.147
Statistical Analysis 212: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 211]; Test type: Superiority; p = 0.8286, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.25 to 0.32], Standard Error of Mean 0.144
Statistical Analysis 213: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3022, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.49 to 0.15], Standard Error of Mean 0.162
Statistical Analysis 214: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 213]; Test type: Superiority; p = 0.8022, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.35 to 0.27], Standard Error of Mean 0.158
Statistical Analysis 215: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5665, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.42 to 0.23], Standard Error of Mean 0.165
Statistical Analysis 216: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 215]; Test type: Superiority; p = 0.8170, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.36 to 0.28], Standard Error of Mean 0.161
Statistical Analysis 217: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0404, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.63 to -0.01], Standard Error of Mean 0.155
Statistical Analysis 218: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 217]; Test type: Superiority; p = 0.3128, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.45 to 0.15], Standard Error of Mean 0.151
Statistical Analysis 219: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2400, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.51 to 0.13], Standard Error of Mean 0.162
Statistical Analysis 220: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 219]; Test type: Superiority; p = 0.4840, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.42 to 0.20], Standard Error of Mean 0.157
Statistical Analysis 221: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7768, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.32 to 0.24], Standard Error of Mean 0.141
Statistical Analysis 222: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 221]; Test type: Superiority; p = 0.7713, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.31 to 0.23], Standard Error of Mean 0.137
Statistical Analysis 223: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0716, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.58 to 0.02], Standard Error of Mean 0.151
Statistical Analysis 224: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 223]; Test type: Superiority; p = 0.4317, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.41 to 0.18], Standard Error of Mean 0.148
Statistical Analysis 225: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2115, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.52 to 0.12], Standard Error of Mean 0.162
Statistical Analysis 226: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 225]; Test type: Superiority; p = 0.2818, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.48 to 0.14], Standard Error of Mean 0.158
Statistical Analysis 227: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2018, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.46 to 0.10], Standard Error of Mean 0.140
Statistical Analysis 228: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 227]; Test type: Superiority; p = 0.6554, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.33 to 0.21], Standard Error of Mean 0.137
Statistical Analysis 229: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4754, MMRM; LS mean difference = 0.12, 95% CI 2-sided [-0.21 to 0.46], Standard Error of Mean 0.168
Statistical Analysis 230: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 229]; Test type: Superiority; p = 0.7776, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.28 to 0.37], Standard Error of Mean 0.163
Statistical Analysis 231: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7172, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.50 to 0.35], Standard Error of Mean 0.213
Statistical Analysis 232: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 231]; Test type: Superiority; p = 0.4791, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.55 to 0.26], Standard Error of Mean 0.203
Statistical Analysis 233: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Agitation, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3562, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.48 to 0.17], Standard Error of Mean 0.164
Statistical Analysis 234: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 233]; Test type: Superiority; p = 0.8859, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.30 to 0.34], Standard Error of Mean 0.162
Statistical Analysis 235: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5888, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.49 to 0.28], Standard Error of Mean 0.192
Statistical Analysis 236: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 235]; Test type: Superiority; p = 0.3992, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.53 to 0.21], Standard Error of Mean 0.187
Statistical Analysis 237: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1212, MMRM; LS mean difference = -0.35, 95% CI 2-sided [-0.80 to 0.10], Standard Error of Mean 0.227
Statistical Analysis 238: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 237]; Test type: Superiority; p = 0.3185, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.66 to 0.22], Standard Error of Mean 0.221
Statistical Analysis 239: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4809, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.62 to 0.29], Standard Error of Mean 0.231
Statistical Analysis 240: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 239]; Test type: Superiority; p = 0.8953, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.42 to 0.48], Standard Error of Mean 0.225
Statistical Analysis 241: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5616, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.57 to 0.31], Standard Error of Mean 0.223
Statistical Analysis 242: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 241]; Test type: Superiority; p = 0.8571, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.39 to 0.47], Standard Error of Mean 0.216
Statistical Analysis 243: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0037, MMRM; LS mean difference = -0.63, 95% CI 2-sided [-1.05 to -0.21], Standard Error of Mean 0.213
Statistical Analysis 244: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 243]; Test type: Superiority; p = 0.0386, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.84 to -0.02], Standard Error of Mean 0.206
Statistical Analysis 245: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0044, MMRM; LS mean difference = -0.63, 95% CI 2-sided [-1.05 to -0.20], Standard Error of Mean 0.216
Statistical Analysis 246: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 245]; Test type: Superiority; p = 0.8308, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.46 to 0.37], Standard Error of Mean 0.208
Statistical Analysis 247: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0388, MMRM; LS mean difference = -0.45, 95% CI 2-sided [-0.87 to -0.02], Standard Error of Mean 0.215
Statistical Analysis 248: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 247]; Test type: Superiority; p = 0.1622, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.71 to 0.12], Standard Error of Mean 0.209
Statistical Analysis 249: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0179, MMRM; LS mean difference = -0.49, 95% CI 2-sided [-0.89 to -0.09], Standard Error of Mean 0.204
Statistical Analysis 250: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 249]; Test type: Superiority; p = 0.4283, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.55 to 0.24], Standard Error of Mean 0.198
Statistical Analysis 251: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1899, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.72 to 0.15], Standard Error of Mean 0.219
Statistical Analysis 252: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 251]; Test type: Superiority; p = 0.8022, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.48 to 0.37], Standard Error of Mean 0.213
Statistical Analysis 253: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3780, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.62 to 0.24], Standard Error of Mean 0.215
Statistical Analysis 254: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 253]; Test type: Superiority; p = 0.8110, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.47 to 0.36], Standard Error of Mean 0.210
Statistical Analysis 255: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8908, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.58 to 0.50], Standard Error of Mean 0.272
Statistical Analysis 256: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 255]; Test type: Superiority; p = 0.3596, MMRM; LS mean difference = 0.24, 95% CI 2-sided [-0.28 to 0.76], Standard Error of Mean 0.263
Statistical Analysis 257: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7617, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.67 to 0.49], Standard Error of Mean 0.293
Statistical Analysis 258: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 257]; Test type: Superiority; p = 0.5498, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.73 to 0.39], Standard Error of Mean 0.281
Statistical Analysis 259: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Psychic, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2066, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.76 to 0.17], Standard Error of Mean 0.235
Statistical Analysis 260: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 259]; Test type: Superiority; p = 0.2321, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.73 to 0.18], Standard Error of Mean 0.230
Statistical Analysis 261: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5582, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.49 to 0.27], Standard Error of Mean 0.191
Statistical Analysis 262: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 261]; Test type: Superiority; p = 0.2945, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.56 to 0.17], Standard Error of Mean 0.186
Statistical Analysis 263: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2684, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.64 to 0.18], Standard Error of Mean 0.208
Statistical Analysis 264: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 263]; Test type: Superiority; p = 0.9396, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.42 to 0.39], Standard Error of Mean 0.202
Statistical Analysis 265: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0283, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.82 to -0.05], Standard Error of Mean 0.195
Statistical Analysis 266: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 265]; Test type: Superiority; p = 0.1794, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.63 to 0.12], Standard Error of Mean 0.189
Statistical Analysis 267: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1091, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.68 to 0.07], Standard Error of Mean 0.188
Statistical Analysis 268: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 267]; Test type: Superiority; p = 0.7921, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.41 to 0.31], Standard Error of Mean 0.182
Statistical Analysis 269: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0055, MMRM; LS mean difference = -0.47, 95% CI 2-sided [-0.80 to -0.14], Standard Error of Mean 0.166
Statistical Analysis 270: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 269]; Test type: Superiority; p = 0.0300, MMRM; LS mean difference = -0.35, 95% CI 2-sided [-0.67 to -0.03], Standard Error of Mean 0.161
Statistical Analysis 271: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0118, MMRM; LS mean difference = -0.47, 95% CI 2-sided [-0.84 to -0.11], Standard Error of Mean 0.185
Statistical Analysis 272: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 271]; Test type: Superiority; p = 0.2266, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.57 to 0.14], Standard Error of Mean 0.178
Statistical Analysis 273: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0025, MMRM; LS mean difference = -0.56, 95% CI 2-sided [-0.92 to -0.20], Standard Error of Mean 0.181
Statistical Analysis 274: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 273]; Test type: Superiority; p = 0.0555, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.69 to 0.01], Standard Error of Mean 0.176
Statistical Analysis 275: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0013, MMRM; LS mean difference = -0.58, 95% CI 2-sided [-0.93 to -0.23], Standard Error of Mean 0.176
Statistical Analysis 276: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 275]; Test type: Superiority; p = 0.0775, MMRM; LS mean difference = -0.31, 95% CI 2-sided [-0.64 to 0.03], Standard Error of Mean 0.171
Statistical Analysis 277: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0006, MMRM; LS mean difference = -0.67, 95% CI 2-sided [-1.05 to -0.30], Standard Error of Mean 0.190
Statistical Analysis 278: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 277]; Test type: Superiority; p = 0.0415, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-0.75 to -0.01], Standard Error of Mean 0.185
Statistical Analysis 279: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0581, MMRM; LS mean difference = -0.37, 95% CI 2-sided [-0.75 to 0.01], Standard Error of Mean 0.193
Statistical Analysis 280: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 279]; Test type: Superiority; p = 0.6826, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.45 to 0.30], Standard Error of Mean 0.188
Statistical Analysis 281: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0912, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-0.83 to 0.06], Standard Error of Mean 0.226
Statistical Analysis 282: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 281]; Test type: Superiority; p = 0.3988, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.62 to 0.25], Standard Error of Mean 0.218
Statistical Analysis 283: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0504, MMRM; LS mean difference = -0.46, 95% CI 2-sided [-0.91 to 0.00], Standard Error of Mean 0.231
Statistical Analysis 284: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 283]; Test type: Superiority; p = 0.6019, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.55 to 0.32], Standard Error of Mean 0.220
Statistical Analysis 285: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Anxiety Somatic, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0070, MMRM; LS mean difference = -0.61, 95% CI 2-sided [-1.05 to -0.17], Standard Error of Mean 0.222
Statistical Analysis 286: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 285]; Test type: Superiority; p = 0.3785, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.62 to 0.24], Standard Error of Mean 0.218
Statistical Analysis 287: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9609, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.32 to 0.31], Standard Error of Mean 0.159
Statistical Analysis 288: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 287]; Test type: Superiority; p = 0.9183, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.32 to 0.29], Standard Error of Mean 0.154
Statistical Analysis 289: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0710, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-0.57 to 0.02], Standard Error of Mean 0.149
Statistical Analysis 290: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 289]; Test type: Superiority; p = 0.2607, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.45 to 0.12], Standard Error of Mean 0.143
Statistical Analysis 291: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2466, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.50 to 0.13], Standard Error of Mean 0.158
Statistical Analysis 292: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 291]; Test type: Superiority; p = 0.3461, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.45 to 0.16], Standard Error of Mean 0.153
Statistical Analysis 293: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0919, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.60 to 0.05], Standard Error of Mean 0.162
Statistical Analysis 294: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 293]; Test type: Superiority; p = 0.7554, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.36 to 0.26], Standard Error of Mean 0.157
Statistical Analysis 295: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0150, MMRM; LS mean difference = -0.41, 95% CI 2-sided [-0.74 to -0.08], Standard Error of Mean 0.166
Statistical Analysis 296: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 295]; Test type: Superiority; p = 0.0482, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.64 to 0.00], Standard Error of Mean 0.160
Statistical Analysis 297: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0003, MMRM; LS mean difference = -0.61, 95% CI 2-sided [-0.93 to -0.28], Standard Error of Mean 0.163
Statistical Analysis 298: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 297]; Test type: Superiority; p = 0.1182, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.56 to 0.06], Standard Error of Mean 0.156
Statistical Analysis 299: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0008, MMRM; LS mean difference = -0.55, 95% CI 2-sided [-0.87 to -0.24], Standard Error of Mean 0.159
Statistical Analysis 300: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 299]; Test type: Superiority; p = 0.1379, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.54 to 0.08], Standard Error of Mean 0.154
Statistical Analysis 301: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0040, MMRM; LS mean difference = -0.43, 95% CI 2-sided [-0.71 to -0.14], Standard Error of Mean 0.145
Statistical Analysis 302: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 301]; Test type: Superiority; p = 0.3100, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.42 to 0.14], Standard Error of Mean 0.140
Statistical Analysis 303: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0003, MMRM; LS mean difference = -0.56, 95% CI 2-sided [-0.85 to -0.26], Standard Error of Mean 0.148
Statistical Analysis 304: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 303]; Test type: Superiority; p = 0.0223, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.61 to -0.05], Standard Error of Mean 0.143
Statistical Analysis 305: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0276, MMRM; LS mean difference = -0.37, 95% CI 2-sided [-0.70 to -0.04], Standard Error of Mean 0.166
Statistical Analysis 306: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 305]; Test type: Superiority; p = 0.8516, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.35 to 0.29], Standard Error of Mean 0.161
Statistical Analysis 307: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1669, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.63 to 0.11], Standard Error of Mean 0.186
Statistical Analysis 308: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 307]; Test type: Superiority; p = 0.4935, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.48 to 0.23], Standard Error of Mean 0.180
Statistical Analysis 309: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0202, MMRM; LS mean difference = -0.47, 95% CI 2-sided [-0.86 to -0.07], Standard Error of Mean 0.197
Statistical Analysis 310: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 309]; Test type: Superiority; p = 0.2683, MMRM; LS mean difference = -0.21, 95% CI 2-sided [-0.58 to 0.16], Standard Error of Mean 0.188
Statistical Analysis 311: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms GI, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0531, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.65 to 0.00], Standard Error of Mean 0.165
Statistical Analysis 312: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 311]; Test type: Superiority; p = 0.5609, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.41 to 0.22], Standard Error of Mean 0.160
Statistical Analysis 313: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6779, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.30 to 0.19], Standard Error of Mean 0.123
Statistical Analysis 314: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 313]; Test type: Superiority; p = 0.4559, MMRM; LS mean difference = 0.09, 95% CI 2-sided [-0.15 to 0.32], Standard Error of Mean 0.119
Statistical Analysis 315: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2254, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.43 to 0.10], Standard Error of Mean 0.133
Statistical Analysis 316: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 315]; Test type: Superiority; p = 0.6437, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.32 to 0.20], Standard Error of Mean 0.129
Statistical Analysis 317: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6678, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.32 to 0.21], Standard Error of Mean 0.133
Statistical Analysis 318: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 317]; Test type: Superiority; p = 0.9321, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.27 to 0.24], Standard Error of Mean 0.129
Statistical Analysis 319: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9778, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.31 to 0.32], Standard Error of Mean 0.157
Statistical Analysis 320: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 319]; Test type: Superiority; p = 0.9307, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.29 to 0.31], Standard Error of Mean 0.152
Statistical Analysis 321: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6791, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.41 to 0.27], Standard Error of Mean 0.172
Statistical Analysis 322: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 321]; Test type: Superiority; p = 0.7769, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.28 to 0.38], Standard Error of Mean 0.167
Statistical Analysis 323: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7206, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.38 to 0.26], Standard Error of Mean 0.163
Statistical Analysis 324: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 323]; Test type: Superiority; p = 0.3549, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.45 to 0.16], Standard Error of Mean 0.156
Statistical Analysis 325: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0231, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-0.70 to -0.05], Standard Error of Mean 0.164
Statistical Analysis 326: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 325]; Test type: Superiority; p = 0.1450, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.55 to 0.08], Standard Error of Mean 0.159
Statistical Analysis 327: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0855, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.60 to 0.04], Standard Error of Mean 0.162
Statistical Analysis 328: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 327]; Test type: Superiority; p = 0.3068, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.47 to 0.15], Standard Error of Mean 0.157
Statistical Analysis 329: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0069, MMRM; LS mean difference = -0.45, 95% CI 2-sided [-0.77 to -0.13], Standard Error of Mean 0.164
Statistical Analysis 330: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 329]; Test type: Superiority; p = 0.2174, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.51 to 0.12], Standard Error of Mean 0.159
Statistical Analysis 331: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1020, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.63 to 0.06], Standard Error of Mean 0.174
Statistical Analysis 332: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 331]; Test type: Superiority; p = 0.9587, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.33 to 0.35], Standard Error of Mean 0.170
Statistical Analysis 333: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1690, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.69 to 0.12], Standard Error of Mean 0.203
Statistical Analysis 334: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 333]; Test type: Superiority; p = 0.7919, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.34 to 0.44], Standard Error of Mean 0.197
Statistical Analysis 335: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0192, MMRM; LS mean difference = -0.49, 95% CI 2-sided [-0.89 to -0.08], Standard Error of Mean 0.205
Statistical Analysis 336: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 335]; Test type: Superiority; p = 0.3887, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.56 to 0.22], Standard Error of Mean 0.196
Statistical Analysis 337: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Somatic Symptoms General, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0719, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.72 to 0.03], Standard Error of Mean 0.189
Statistical Analysis 338: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 337]; Test type: Superiority; p = 0.1195, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.66 to 0.08], Standard Error of Mean 0.185
Statistical Analysis 339: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9552, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.16 to 0.15], Standard Error of Mean 0.079
Statistical Analysis 340: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 339]; Test type: Superiority; p = 0.0384, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.31 to -0.01], Standard Error of Mean 0.076
Statistical Analysis 341: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2582, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.30 to 0.08], Standard Error of Mean 0.097
Statistical Analysis 342: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 341]; Test type: Superiority; p = 0.1511, MMRM; LS mean difference = -0.14, 95% CI 2-sided [-0.32 to 0.05], Standard Error of Mean 0.094
Statistical Analysis 343: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4631, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.34 to 0.16], Standard Error of Mean 0.126
Statistical Analysis 344: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 343]; Test type: Superiority; p = 0.4628, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.33 to 0.15], Standard Error of Mean 0.123
Statistical Analysis 345: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9005, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.23 to 0.20], Standard Error of Mean 0.110
Statistical Analysis 346: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 345]; Test type: Superiority; p = 0.1121, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.38 to 0.04], Standard Error of Mean 0.107
Statistical Analysis 347: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4167, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.40 to 0.17], Standard Error of Mean 0.145
Statistical Analysis 348: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 347]; Test type: Superiority; p = 0.4071, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.40 to 0.16], Standard Error of Mean 0.141
Statistical Analysis 349: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1278, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-0.53 to 0.07], Standard Error of Mean 0.150
Statistical Analysis 350: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 349]; Test type: Superiority; p = 0.0573, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.57 to 0.01], Standard Error of Mean 0.145
Statistical Analysis 351: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4842, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.42 to 0.20], Standard Error of Mean 0.156
Statistical Analysis 352: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 351]; Test type: Superiority; p = 0.0692, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.58 to 0.02], Standard Error of Mean 0.152
Statistical Analysis 353: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4028, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.44 to 0.18], Standard Error of Mean 0.157
Statistical Analysis 354: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 353]; Test type: Superiority; p = 0.0354, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.63 to -0.02], Standard Error of Mean 0.154
Statistical Analysis 355: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1228, MMRM; LS mean difference = -0.24, 95% CI 2-sided [-0.55 to 0.07], Standard Error of Mean 0.156
Statistical Analysis 356: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 355]; Test type: Superiority; p = 0.0099, MMRM; LS mean difference = -0.40, 95% CI 2-sided [-0.70 to -0.10], Standard Error of Mean 0.152
Statistical Analysis 357: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2174, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.53 to 0.12], Standard Error of Mean 0.164
Statistical Analysis 358: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 357]; Test type: Superiority; p = 0.0820, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-0.60 to 0.04], Standard Error of Mean 0.161
Statistical Analysis 359: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2642, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.60 to 0.17], Standard Error of Mean 0.194
Statistical Analysis 360: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 359]; Test type: Superiority; p = 0.0718, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.72 to 0.03], Standard Error of Mean 0.189
Statistical Analysis 361: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3055, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.64 to 0.20], Standard Error of Mean 0.212
Statistical Analysis 362: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 361]; Test type: Superiority; p = 0.3533, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.59 to 0.21], Standard Error of Mean 0.202
Statistical Analysis 363: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Genital Symptoms, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4514, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.53 to 0.24], Standard Error of Mean 0.193
Statistical Analysis 364: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 363]; Test type: Superiority; p = 0.4907, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.51 to 0.25], Standard Error of Mean 0.191
Statistical Analysis 365: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6949, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.36 to 0.24], Standard Error of Mean 0.151
Statistical Analysis 366: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 365]; Test type: Superiority; p = 0.4670, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.40 to 0.18], Standard Error of Mean 0.147
Statistical Analysis 367: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6556, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-0.39 to 0.25], Standard Error of Mean 0.160
Statistical Analysis 368: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 367]; Test type: Superiority; p = 0.9272, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.32 to 0.29], Standard Error of Mean 0.156
Statistical Analysis 369: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1395, MMRM; LS mean difference = -0.24, 95% CI 2-sided [-0.57 to 0.08], Standard Error of Mean 0.164
Statistical Analysis 370: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 369]; Test type: Superiority; p = 0.2601, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-0.50 to 0.14], Standard Error of Mean 0.159
Statistical Analysis 371: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5626, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.40 to 0.22], Standard Error of Mean 0.158
Statistical Analysis 372: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 371]; Test type: Superiority; p = 0.4622, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.42 to 0.19], Standard Error of Mean 0.153
Statistical Analysis 373: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2858, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.46 to 0.14], Standard Error of Mean 0.151
Statistical Analysis 374: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 373]; Test type: Superiority; p = 0.5369, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.38 to 0.20], Standard Error of Mean 0.146
Statistical Analysis 375: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1510, MMRM; LS mean difference = -0.22, 95% CI 2-sided [-0.52 to 0.08], Standard Error of Mean 0.150
Statistical Analysis 376: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 375]; Test type: Superiority; p = 0.5107, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.38 to 0.19], Standard Error of Mean 0.146
Statistical Analysis 377: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3301, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.45 to 0.15], Standard Error of Mean 0.151
Statistical Analysis 378: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 377]; Test type: Superiority; p = 0.5139, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.39 to 0.19], Standard Error of Mean 0.147
Statistical Analysis 379: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4073, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.40 to 0.17], Standard Error of Mean 0.144
Statistical Analysis 380: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 379]; Test type: Superiority; p = 0.4649, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.38 to 0.17], Standard Error of Mean 0.140
Statistical Analysis 381: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6926, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.34 to 0.22], Standard Error of Mean 0.141
Statistical Analysis 382: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 381]; Test type: Superiority; p = 0.7260, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.22 to 0.32], Standard Error of Mean 0.137
Statistical Analysis 383: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1486, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.47 to 0.07], Standard Error of Mean 0.136
Statistical Analysis 384: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 383]; Test type: Superiority; p = 0.4800, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.36 to 0.17], Standard Error of Mean 0.133
Statistical Analysis 385: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7792, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.40 to 0.30], Standard Error of Mean 0.177
Statistical Analysis 386: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 385]; Test type: Superiority; p = 0.8644, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.31 to 0.37], Standard Error of Mean 0.171
Statistical Analysis 387: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7994, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.27 to 0.35], Standard Error of Mean 0.158
Statistical Analysis 388: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 387]; Test type: Superiority; p = 0.0811, MMRM; LS mean difference = 0.27, 95% CI 2-sided [-0.03 to 0.57], Standard Error of Mean 0.152
Statistical Analysis 389: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hypochondriasis, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6978, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.34 to 0.23], Standard Error of Mean 0.144
Statistical Analysis 390: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 389]; Test type: Superiority; p = 0.9749, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.28 to 0.28], Standard Error of Mean 0.141
Statistical Analysis 391: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3158, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.08 to 0.24], Standard Error of Mean 0.081
Statistical Analysis 392: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 391]; Test type: Superiority; p = 0.1901, MMRM; LS mean difference = 0.10, 95% CI 2-sided [-0.05 to 0.26], Standard Error of Mean 0.079
Statistical Analysis 393: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7229, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.12 to 0.17], Standard Error of Mean 0.073
Statistical Analysis 394: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 393]; Test type: Superiority; p = 0.2715, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-0.06 to 0.22], Standard Error of Mean 0.071
Statistical Analysis 395: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5421, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.12 to 0.22], Standard Error of Mean 0.086
Statistical Analysis 396: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 395]; Test type: Superiority; p = 0.7215, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.14 to 0.19], Standard Error of Mean 0.083
Statistical Analysis 397: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2246, MMRM; LS mean difference = 0.12, 95% CI 2-sided [-0.07 to 0.31], Standard Error of Mean 0.098
Statistical Analysis 398: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 397]; Test type: Superiority; p = 0.9671, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.19 to 0.19], Standard Error of Mean 0.096
Statistical Analysis 399: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6527, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.29 to 0.19], Standard Error of Mean 0.121
Statistical Analysis 400: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 399]; Test type: Superiority; p = 0.1647, MMRM; LS mean difference = -0.17, 95% CI 2-sided [-0.40 to 0.07], Standard Error of Mean 0.118
Statistical Analysis 401: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7093, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-0.18 to 0.26], Standard Error of Mean 0.110
Statistical Analysis 402: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 401]; Test type: Superiority; p = 0.6333, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.26 to 0.16], Standard Error of Mean 0.107
Statistical Analysis 403: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5238, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.31 to 0.16], Standard Error of Mean 0.120
Statistical Analysis 404: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 403]; Test type: Superiority; p = 0.0782, MMRM; LS mean difference = -0.21, 95% CI 2-sided [-0.44 to 0.02], Standard Error of Mean 0.117
Statistical Analysis 405: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2346, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.44 to 0.11], Standard Error of Mean 0.138
Statistical Analysis 406: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 405]; Test type: Superiority; p = 0.0631, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-0.52 to 0.01], Standard Error of Mean 0.134
Statistical Analysis 407: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6274, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.32 to 0.20], Standard Error of Mean 0.131
Statistical Analysis 408: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 407]; Test type: Superiority; p = 0.3589, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.37 to 0.14], Standard Error of Mean 0.128
Statistical Analysis 409: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7604, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.43 to 0.31], Standard Error of Mean 0.187
Statistical Analysis 410: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 409]; Test type: Superiority; p = 0.1106, MMRM; LS mean difference = -0.30, 95% CI 2-sided [-0.66 to 0.07], Standard Error of Mean 0.185
Statistical Analysis 411: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9776, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.43 to 0.45], Standard Error of Mean 0.222
Statistical Analysis 412: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 411]; Test type: Superiority; p = 0.3239, MMRM; LS mean difference = -0.21, 95% CI 2-sided [-0.65 to 0.22], Standard Error of Mean 0.217
Statistical Analysis 413: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6736, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.57 to 0.37], Standard Error of Mean 0.238
Statistical Analysis 414: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 413]; Test type: Superiority; p = 0.6136, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.58 to 0.34], Standard Error of Mean 0.231
Statistical Analysis 415: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Loss of Weight, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1141, MMRM; LS mean difference = -0.31, 95% CI 2-sided [-0.70 to 0.08], Standard Error of Mean 0.195
Statistical Analysis 416: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 415]; Test type: Superiority; p = 0.2185, MMRM; LS mean difference = -0.24, 95% CI 2-sided [-0.62 to 0.14], Standard Error of Mean 0.194
Statistical Analysis 417: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6191, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.08 to 0.13], Standard Error of Mean 0.054
Statistical Analysis 418: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 417]; Test type: Superiority; p = 0.6169, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.08 to 0.13], Standard Error of Mean 0.053
Statistical Analysis 419: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9911, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.054
Statistical Analysis 420: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 419]; Test type: Superiority; p = 0.3360, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.05 to 0.15], Standard Error of Mean 0.053
Statistical Analysis 421: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9638, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.054
Statistical Analysis 422: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 421]; Test type: Superiority; p = 0.1610, MMRM; LS mean difference = 0.07, 95% CI 2-sided [-0.03 to 0.18], Standard Error of Mean 0.053
Statistical Analysis 423: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5763, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.14 to 0.08], Standard Error of Mean 0.054
Statistical Analysis 424: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 423]; Test type: Superiority; p = 0.0599, MMRM; LS mean difference = 0.10, 95% CI 2-sided [0.00 to 0.20], Standard Error of Mean 0.053
Statistical Analysis 425: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3916, MMRM; LS mean difference = -0.05, 95% CI 2-sided [-0.15 to 0.06], Standard Error of Mean 0.054
Statistical Analysis 426: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 425]; Test type: Superiority; p = 0.9602, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.10 to 0.11], Standard Error of Mean 0.053
Statistical Analysis 427: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9676, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.11 to 0.11], Standard Error of Mean 0.055
Statistical Analysis 428: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 427]; Test type: Superiority; p = 0.6397, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.08 to 0.13], Standard Error of Mean 0.053
Statistical Analysis 429: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3400, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.05 to 0.16], Standard Error of Mean 0.054
Statistical Analysis 430: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 429]; Test type: Superiority; p = 0.3472, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.05 to 0.15], Standard Error of Mean 0.053
Statistical Analysis 431: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9160, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.054
Statistical Analysis 432: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 431]; Test type: Superiority; p = 0.5948, MMRM; LS mean difference = -0.03, 95% CI 2-sided [-0.13 to 0.08], Standard Error of Mean 0.053
Statistical Analysis 433: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3755, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.06 to 0.16], Standard Error of Mean 0.054
Statistical Analysis 434: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 433]; Test type: Superiority; p = 0.9752, MMRM; LS mean difference = 0.00, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.053
Statistical Analysis 435: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9188, MMRM; LS mean difference = -0.01, 95% CI 2-sided [-0.11 to 0.10], Standard Error of Mean 0.054
Statistical Analysis 436: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 435]; Test type: Superiority; p = 0.6379, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.08 to 0.13], Standard Error of Mean 0.053
Statistical Analysis 437: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4967, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.16 to 0.08], Standard Error of Mean 0.061
Statistical Analysis 438: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 437]; Test type: Superiority; p = 0.3492, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.17 to 0.06], Standard Error of Mean 0.059
Statistical Analysis 439: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7136, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.10 to 0.14], Standard Error of Mean 0.062
Statistical Analysis 440: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 439]; Test type: Superiority; p = 0.8163, MMRM; LS mean difference = 0.01, 95% CI 2-sided [-0.10 to 0.13], Standard Error of Mean 0.059
Statistical Analysis 441: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Insight, Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2825, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-0.17 to 0.05], Standard Error of Mean 0.055
Statistical Analysis 442: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 7, analysis 441]; Test type: Superiority; p = 0.1603, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.18 to 0.03], Standard Error of Mean 0.054

8. Secondary Outcome: Change From Baseline at Key Time Points in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicates more severe depression. A negative change from baseline indicates less severe depression. A positive change from baseline indicates more severe depression.
Time Frame: Baseline, Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
score on a scale
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | -19.98 (1.688) | -26.84 (1.822) | -24.19 (1.797)
  Day 7: number analyzed (Participants) | 43 | 38 | 39
  Day 7 | -19.01 (1.865) | -23.31 (2.001) | -20.32 (1.982)
  Day 30: number analyzed (Participants) | 42 | 35 | 36
  Day 30 | -19.43 (1.917) | -25.06 (2.091) | -23.02 (2.080)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 60: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0054, MMRM; LS mean difference = -6.85, 95% CI 2-sided [-11.64 to -2.07], Standard Error of Mean 2.414
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0763, MMRM; LS mean difference = -4.20, 95% CI 2-sided [-8.86 to 0.45], Standard Error of Mean 2.350
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1101, MMRM; LS mean difference = -4.30, 95% CI 2-sided [-9.60 to 0.99], Standard Error of Mean 2.673
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.6167, MMRM; LS mean difference = -1.31, 95% CI 2-sided [-6.50 to 3.87], Standard Error of Mean 2.618
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 30: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0447, MMRM; LS mean difference = -5.64, 95% CI 2-sided [-11.14 to -0.14], Standard Error of Mean 2.777
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.1908, MMRM; LS mean difference = -3.59, 95% CI 2-sided [-8.99 to 1.81], Standard Error of Mean 2.726

9. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response
Description: The CGI-I item employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions. CGI-I response was defined as having a score of 1 (very much improved) or 2 (much improved).
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
percentage of participants
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | 55.8 | 83.8 | 82.1
  Day 7: number analyzed (Participants) | 43 | 38 | 39
  Day 7 | 46.5 | 71.1 | 64.1
  Day 30: number analyzed (Participants) | 42 | 35 | 36
  Day 30 | 52.4 | 80.0 | 72.2
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Hour 60: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0131, GEE method; Odds Ratio (OR) = 4.0, 95% CI 2-sided [1.3 to 11.7]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0095, GEE method; Odds Ratio (OR) = 4.0, 95% CI 2-sided [1.4 to 11.6]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Day 7: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0323, GEE method; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.1 to 7.5]
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.0931, GEE method; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.9 to 5.3]
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Day 30: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0139, GEE method; Odds Ratio (OR) = 3.6, 95% CI 2-sided [1.3 to 10.0]
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 9, analysis 5]; Test type: Superiority; p = 0.0460, GEE method; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.0 to 6.9]

10. Secondary Outcome: Change From Baseline in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) Total Score
Description: The GAD-7 is a participant-rated, generalized anxiety symptom severity scale. Scoring for GAD-7 generalized anxiety is calculated by assigning scores of 0 = "not at all sure," 1 = "several days," 2 = "over half the days," and 3 = "nearly every day" to the response categories. The GAD-7 total score for the seven items ranges from 0 to 21, where a score of 0 to 4 = minimal anxiety, 5 to 9 = mild anxiety, 10 to 14 = moderate anxiety, and 15 to 21 = severe anxiety. The GAD-7 total score was calculated as the sum of the seven individual item scores. A negative change from baseline indicates less anxiety. A positive change from baseline indicates more anxiety.
Time Frame: Baseline, Hour 60, Days 7, 14, 21 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
score on a scale
  Hour 60: number analyzed (Participants) | 43 | 37 | 39
  Hour 60 | -6.95 (1.012) | -8.08 (1.095) | -7.99 (1.087)
  Day 7: number analyzed (Participants) | 43 | 37 | 38
  Day 7 | -6.57 (0.947) | -9.13 (1.025) | -6.32 (1.034)
  Day 14: number analyzed (Participants) | 30 | 22 | 25
  Day 14 | -8.60 (1.081) | -9.20 (1.210) | -8.71 (1.191)
  Day 21: number analyzed (Participants) | 30 | 22 | 26
  Day 21 | -8.47 (1.093) | -8.53 (1.224) | -9.22 (1.199)
  Day 30: number analyzed (Participants) | 42 | 34 | 35
  Day 30 | -7.70 (1.023) | -9.72 (1.129) | -9.15 (1.135)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Hour 60: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4389, MMRM; LS mean difference = -1.13, 95% CI 2-sided [-4.01 to 1.75], Standard Error of Mean 1.454
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.4645, MMRM; LS mean difference = -1.05, 95% CI 2-sided [-3.88 to 1.78], Standard Error of Mean 1.427
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 7: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0622, MMRM; LS mean difference = -2.56, 95% CI 2-sided [-5.24 to 0.13], Standard Error of Mean 1.356
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 10, analysis 3]; Test type: Superiority; p = 0.8495, MMRM; LS mean difference = 0.25, 95% CI 2-sided [-2.40 to 2.91], Standard Error of Mean 1.338
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 14: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7063, MMRM; LS mean difference = -0.60, 95% CI 2-sided [-3.75 to 2.55], Standard Error of Mean 1.590
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.9434, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-3.19 to 2.97], Standard Error of Mean 1.552
Statistical Analysis 7: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 21: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9701, MMRM; LS mean difference = -0.06, 95% CI 2-sided [-3.25 to 3.13], Standard Error of Mean 1.608
Statistical Analysis 8: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.6307, MMRM; LS mean difference = -0.76, 95% CI 2-sided [-3.86 to 2.35], Standard Error of Mean 1.566
Statistical Analysis 9: Comparison: Placebo vs SAGE-547 60 μg/kg/h; Change at Day 30: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1767, MMRM; LS mean difference = -2.02, 95% CI 2-sided [-4.97 to 0.93], Standard Error of Mean 1.488
Statistical Analysis 10: Comparison: Placebo vs SAGE-547 90 μg/kg/h; [analysis description as in outcome 10, analysis 9]; Test type: Superiority; p = 0.3236, MMRM; LS mean difference = -1.46, 95% CI 2-sided [-4.37 to 1.45], Standard Error of Mean 1.468

11. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent AE (TEAE) is defined as an AE with onset on or after the start of study drug infusion, or any worsening of a pre-existing medical condition/AE with onset on or after the start of study drug infusion.
Time Frame: Up to approximately 37 days.
Population: The Safety Set included all randomized participants who started the study drug infusion.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
percentage of participants | 51.2 | 50.0 | 53.7

12. Secondary Outcome: Time to Change in Antidepressant Medication
Description: The time to first start or increase in the dose and time to first stop or decrease in the dose of any antidepressant medication.
Time Frame: Up to approximately 37 days.
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 43 | 38 | 41
days
  Time to first start/increase in dose: number analyzed (Participants) | 3 | 4 | 5
  Time to first start/increase in dose | 16 [5 to 22] | 12 [5 to 34] | 8 [4 to 29]
  Time to first stop/decrease in dose: number analyzed (Participants) | 0 | 1 | 1
  Time to first stop/decrease in dose |  | 29 [29 to 29] | 19 [19 to 19]

ADVERSE EVENTS:
Time Frame: Up to approximately 37 days.
Description: The Safety Set included all randomized participants who started the study drug infusion.
Arm/Group | Placebo | SAGE-547 60 μg/kg/h | SAGE-547 90 μg/kg/h
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/38 | 0/41
Other Adverse Events (participants affected / at risk) | 9/43 | 17/38 | 13/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-547 60 μg/kg/h (N=38) | SAGE-547 90 μg/kg/h (N=41)
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | SAGE-547 60 μg/kg/h (N=38) | SAGE-547 90 μg/kg/h (N=41)
Dry mouth (Gastrointestinal disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 0
Infusion site pain (General disorders) | 1 | 1 | 4
Dizziness (Nervous system disorders) | 1 | 6 | 6
Headache (Nervous system disorders) | 7 | 7 | 6
Loss of consciousness (Nervous system disorders) | 0 | 2 | 1
Somnolence (Nervous system disorders) | 3 | 7 | 2
Flushing (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02942004/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT02942004/SAP_001.pdf